## GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | ÷ | Reporting and Analysis Plan for Study 201283: An Exploratory Study to Investigate the Use of Biotelemetry to Identify Markers of Disease Progression in Subjects with Amyotrophic Lateral Sclerosis |
|---|---|---|
| <b>Compound Number</b> | : | Non-compound |
| <b>Effective Date</b> | | 03-AUG-2017 |

# **Description:**

The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol [GlaxoSmithKline Document Number 2014N211002\_00] and Protocol amendment [GlaxoSmithKline Document Number 2014N211002\_02].

This RAP is intended to describe the exploratory and safety analyses required for the study.

This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### **Author's Name and Functional Area:**

| PPD | 02 AUC 2017 |
|------------------------------|-------------|
| Associate Statistician (QSI) | 03-AUG-2017 |
| PPD | 03-AUG-2017 |
| Principal Statistician | 03-A0G-201/ |

#### Approved by:

| PPD | 03-AUG-2017 |
|--------------------------------|-------------|
| Associate Director, Statistics | 03-AUG-2017 |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | REPO | ORTING & ANALYSIS PLAN SYNOPSIS | 4 |
| 2. | SUMN<br>2.1.<br>2.2.<br>2.3. | MARY OF KEY PROTOCOL INFORMATION | 6 |
| | 2.4. | Statistical Hypotheses | |
| 3. | PLANI<br>3.1.<br>3.2. | NED ANALYSES | 9 |
| 4. | | Final Analyses YSIS POPULATIONS | |
| т. | 4.1. | Protocol Deviations | |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING<br>/ENTIONS | 11 |
| 6. | STUD | Y POPULATION ANALYSES | 12 |
| | 6.1. | Overview of Planned Analyses | |
| 7. | STATI<br>7.1. | ISTICAL ANALYSESExploratory Analyses | |
| | | <ul><li>7.1.1. Overview of Planned Exploratory Analyses</li><li>7.1.2. Planned Statistical Exploratory Analyses</li></ul> | |
| | 7.2. | Safety Analyses | |
| 8. | REFE | RENCES | 22 |
| 9. | APPE<br>9.1. | NDICESAppendix 1: Time & Events | |
| | J. 1. | 9.1.1. Protocol Defined Time & Events | |
| | 9.2. | Appendix 2: Study States and Phases | |
| | | 9.2.1. Treatment States for AE Data | |
| | 9.3. | Appendix 3: Data Display Standards & Handling Conventions | |
| | | <ul><li>9.3.1. Study Treatment &amp; Sub-group Display Descriptors</li><li>9.3.2. Baseline Definition &amp; Derivations</li></ul> | |
| | | 9.3.2.1 Baseline Definitions | |
| | | 9.3.2.2. Derivations and Handling of Missing Baseline Data | |
| | | 9.3.3. Reporting Process & Standards | |
| | 9.4. | Appendix 4: Derived and Transformed Data | |
| | | 9.4.1. General | |
| | | 9.4.2. Study Population | |
| | | 9.4.3. Exploratory | |
| | 9.5. | Appendix 5: Premature Withdrawals & Handling of Missing Data | |
| | | 9.5.1. Premature Withdrawals | |
| | | 9.5.2. Handling of Missing Data | 31 |

# **CONFIDENTIAL**

| | | 9.5.2.1. | Handling of Par | rtial Dates | <br> | 37 |
|---|---|---|---|---|---|---|
| 9.6. | Appendi | | ntre Studies | | | |
| 9.7. | | | ation of Covaria | | | |
| | 9.7.1. | | f Covariates, Sเ | | | |
| 9.8. | Appendi | x 8: Multiple | Comparisons 8 | & Multiplicity | <br> | 40 |
| 9.9. | | | hecking and Di | | | |
| | Analyse | 3 | | | <br> | 41 |
| | 9.9.1. | Statistical A | Analysis Assum | ptions | <br> | 41 |
| 9.10. | Appendi | x 10: – Abbr | eviations & Tra | de Marks | <br> | 42 |
| | 9.10.1. | Abbreviation | ns | | <br> | 42 |
| | 9.10.2. | Trademark | s | | <br> | 43 |
| 9.11. | Appendi | x 11: List of | Data Displays | | <br> | 44 |
| | 9.11.1. | Data Displa | ay Numbering | | <br> | 44 |
| | 9.11.2. | Mock Exan | nple Shell Refer | rencing | <br> | 44 |
| | 9.11.3. | Study Popu | ulation Tables | | <br> | 45 |
| | 9.11.4. | Exploratory | / Tables | | <br> | . 46 |
| | 9.11.5. | Exploratory | / Figures | | <br> | 63 |
| | 9.11.6. | Safety Tab | les | | <br> | 74 |
| | 9.11.7. | ICH Listing | s | | <br> | 75 |
| | 9.11.8. | Non-ICH Li | istings | | <br> | 77 |

# 1. REPORTING & ANALYSIS PLAN SYNOPSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | The purpose of this reporting and analysis plan (RAP) is to describe all planned analyses and output requirements during the study. |
| Protocol | This RAP is based on the original protocol / protocol amendment 2[(Dated: 21/09/2015) of study MID201283(GSK Document No.: 2014N211002_02] and eCRF Version 3. |
| Primary<br>Objective | There is no primary objective/endpoints in this protocol. See Section 2.2 for exploratory objectives/endpoints. |
| Primary<br>Endpoint | There is no primary objective/endpoints in this protocol. See Section 2.2 for exploratory objectives/endpoints. |
| Study<br>Design | An exploratory, non-controlled, non-drug study in ALS patients. The study consists of two phases: |
| | <ol> <li>A variable length Pilot Phase to test and confirm the algorithms are<br/>capturing movement/physical activity, ensure the data transfer device is<br/>working correctly, and understand the reliability and ease of<br/>use/acceptance of the accelerometer and electrode.</li> </ol> |
| | <ol> <li>A 48-week Core Study Phase to evaluate how measures of<br/>movement/physical activity, speech and HRV relate to ALS disease<br/>progression.</li> </ol> |
| Planned<br>Analyses | A hierarchical approach will be used to focus the analysis on the endpoints where a correlation with either the ALSFRS-R or FVC (as applicable) is present. To begin with, the correlation between the following endpoints will be explored using the analysis method detailed below: |
| | The absolute and change from baseline in the movement/physical activity endpoints as measured by the accelerometer device and the change from baseline in the ALSFRS-R |
| | The absolute and change from baseline in the heart rate variability endpoints as measured by the electrode device and the absolute and change from baseline in the ALSFRS-R |
| | The absolute and change from baseline in the speech endpoints and the absolute and change from baseline in the ALSFRS-R |
| | The absolute and change from baseline in the speech endpoints and the absolute and change from baseline in the FVC |
| | If there's correlation between these endpoints, then further analyses as described in Section 9.7 will be carried out as part of adhoc. |
| Analysis<br>Populations | Enrolled population: This will consist of all subjects who have signed consent and are not a screen failure. |
| | Full Analysis Set (FAS): This will consist of all subjects with at least one post baseline measure for the ALSFRS-R and at least one physical |

# CONFIDENTIAL

| Overview | Key Elements of the RAP |
|---|---|
| | activity/movement measure, night time rest, Heart Rate Variability or Speech assessment endpoint. |
| | Safety: Comprise of all subjects who carried out at least one protocol specified procedure. |
| | Screen Failure: Comprise of all subjects who were a screen failure |
| Hypothesis | The study is designed to explore if there is a relationship between change from baseline in the physical activity/movement, night time rest, heart rate variabil and speech endpoints and change from baseline in the gold standard measure of function (ALSFRS-R and FVC). |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol.

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Exploratory Objectives | Exploratory Endpoints |
| Explore the application of actigraphy: • For measuring movement/physical activity in ALS subjects • As a marker of ALS disease progression | <ul> <li>Change over time in measurements of movement/physical activity by accelerometer reported by day and night time. Measurements include Duration of wear time, (combining day 8 night values to give Wear time), Overall time spen active, Overall time spent sedentary not lying Overall time spent lying, Overall time spent sedentary, Time spent with Sensor off, Total Activity Score, the maximum score from a 1 min window in a 24-hour period and 5 x Active Periods (5 categories &gt;1 to &lt;=2min active up to &gt;30mins active)</li> <li>Change over time in measurements of night time result by accelerometer reported endpoints: Percent Time Lying Down (at night), Number Night Time Movement Episodes, Number Night Time Movement Episodes/Hr, Percent Time Night-time Resulting Efficiency, Rest Fragmentation Index = Move Time/Num Movement Episode, Average Duration Movement Episodes</li> <li>Relationship between the ALSFRS and</li> </ul> |
| | accelerometer measures of movement/activity and night time rest endpoints. |
| Explore the application of continuous remote monitoring of heart rate measures: • For measuring autonomic nervous system function in ALS subjects • As a marker of ALS disease progression | <ul> <li>Change over time in heart rate variability (HRV) as measured by a heartbeat sensing electrode. Measurements include:</li></ul> |

| Objectives | Endpoints |
|---|---|
| | Relationship between the ALSFRS and biotelemetry measures of HRV. |
| Explore the application of digital, quantitative speech testing: • For measuring speech quality in ALS subjects • As a marker of ALS disease progression. | Change over time in digital speech measures of vowel, running speech and word measurements as captured by a high fidelity, acoustic sound capture interface. Measurements include: central tendency of fundamental frequency, jitter, shimmer, maximum gap between words, speaking rate, average phoneme rate, maximum phonation time and % pause time |
| | Relationship between the ALSFRS and digital measures of speech. |
| | <ul> <li>Relationship between Forced Vital Capacity (FVC)<br/>and digital measures of speech.</li> </ul> |
| Explore the impact of the accelerometer and electrode devices on everyday life in subjects with ALS | Subject/caregiver feedback. Feedback may include but not be limited to: comfort of the devices, ease of applying the devices, and ease of data transmission process. |
| Explore the feasibility of biotelemetry transmission of movement/physical activity and HRV data. | Assessed by successful data transmission from the telecommunications hub (Life Insight) to the central secure server at McLaren Applied Technologies (MAT). |
| Safety Objectives | Safety Endpoints |
| Monitor safety and tolerability. | <ul> <li>Type and incidence of adverse events (AEs)<br/>secondary to the devices used in this study.</li> </ul> |
| | <ul> <li>Type and incidence of AEs due to study procedures.</li> </ul> |

# 2.3. Study Design



progression. During this phase, subjects will attend 5 clinic visits to perform gold standard measures of function and perform a series of set

| Overview of Study Design and Key Features | |
|---|---|
| | reference tasks while wearing the accelerometer and electrode. Subjects will also continuously wear the accelerometer and electrode in their routine home-life setting for approximately 3 days after the clinic visits (i.e., home monitoring). In between clinic visits, subjects will attach the accelerometer and electrode and wear it for approximately 3 days in their home. A telephone contact with the subject will be made by the site at the end of each 3-day home monitoring period. |
| Dosing | • NA |
| Treatment<br>Assignment | <ul> <li>This study doesn't include any treatment</li> <li>Treatment of enrolled subjects will be consistent with local standard of clinical care for ALS patients</li> </ul> |
| Interim Analysis | No formal interim analyses will be performed |

# 2.4. Statistical Hypotheses

The study is designed to explore if there is a relationship between change from baseline in the physical activity/movement, heart rate and speech endpoints and change from baseline in the gold standard measures of function (ALSFRS-R and FVC).

#### 3. PLANNED ANALYSES

# 3.1. Interim Analyses

No formal interim analyses will be performed. Review of in stream data will be carried out to understand the utility of the measures and algorithms, the functionality of the data transmission process, and the durability and ease of use/acceptance of the selected accelerometer and electrode. Generated data may result in modifications to the study, such as: changes to the devices/equipment; repositioning of the accelerometer/electrode; modification to the algorithms, the supportive data collection plan or the data transmission process; dropping measures/tests which are not achievable.

McLaren Applied Technologies will not have access to the ALSFRS-R or FVC data and so modifications to the algorithms will be based solely on data collected from the accelerometer/ speech device. All modifications to the algorithms will be documented and version controlled

# 3.2. Final Analyses

The final planned exploratory analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

# 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Enrolled | Comprise of all subjects who have signed consent and are not a screen failure | Study population |
| Full Analysis Set<br>(FAS) | This will consist of all subjects with at least one post baseline measure for the ALSFRS-R and at least one physical activity/movement measure. | <ul><li>Study Population</li><li>Exploratory</li></ul> |
| Safety | Comprise of all subjects who carried out at least one protocol specified procedure. | Safety |
| Screen Failure | Comprise of all subjects who were a screen failure | Study Population |

#### NOTES:

 Please refer to Appendix 11: List of Data Displays which details the population to be used for each displays being generated.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, subject management or subject assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 9.1 | Appendix 1: Time & Events |
| 9.2 | Appendix 2: Treatment States and Phases |
| 9.3 | Appendix 3: Data Display Standards & Handling Conventions |
| 9.4 | Appendix 4: Derived and Transformed Data |
| 9.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| 9.6 | Appendix 6: Multicenter Studies |
| 9.7 | Appendix 7: Examination of Covariates, Subgroups & Other Strata |
| 9.8 | Appendix 8: Multiple Comparisons & Multiplicity |
| 9.9 | Appendix 9: Model Checking and Diagnostics for Statistical Analyses. |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the "Enrolled" OR "FAS" population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

 Table 2
 Overview of Planned Study Population Analyses

| Endpoint / Parameter / Display Type | Data | Displays Gene | erated |
|---|---|---|---|
| | Table | Figure | Listing |
| Subject Disposition | <u>.</u> | | |
| Subject Disposition | Y | | |
| Reasons for Screen Failure | Y | | Y |
| Reasons for Subject Withdrawal | | | Y |
| Subjects by Country and Centre | Y | | |
| Protocol Deviations | · | | |
| Important Protocol Deviations | Y | | Y |
| Subjects with Inclusion/Exclusion Criteria Deviations | | | Υ [1] |
| Populations Analysed | | | |
| Study Populations and Exclusions | Y | | |
| Subjects Excluded from Any Population | | | Υ |
| Demographic and Baseline Characteristics | | | |
| Demographic Characteristics | Y | | Υ |
| Race and Racial Combinations | Y | | Y [2] |
| Medical Conditions and Concomitant Medications | | | |
| Medical Conditions | | | Υ |
| Concomitant Medications | Y | | Y |

# NOTES:

<sup>•</sup> Y = Yes display generated.

<sup>[1]</sup> Listing also includes analysis population exclusions.

<sup>[2]</sup> Listing of race.

# 7. STATISTICAL ANALYSES

# 7.1. Exploratory Analyses

# 7.1.1. Overview of Planned Exploratory Analyses

The efficacy analyses will be based on the "Full Analysis Set" population, unless otherwise specified.

Data Quality Deviators (for data points at each protocol time point):

## Activity & Night time Rest endpoints

For all the actigraphy endpoints if the difference between visits of ALSFRS and Actigraphy is more than 21 days then the data will be excluded and will not be used for the summaries. If the first time point within a visit falls within the 21 days window, then all the time points will be considered.

Using the default sleep times for this study (22:00-07:00) which are derived from the day and night anchor times (set by the day/night algorithms used in this study), the amount of data present for a 24-hour recording period was calculated by adding up the durations for activity classifiers: active + sedentary [where sedentary = sedentary not lying + lying]. If the amount of data present is too low (conversely the amount of "off" time is too high) then the data will not be representative of a full day or night, because a subject's pattern of activity throughout a day or night is not expected to be homogenous or uniform.

A review of the literature showed that a variety of rules can be used, ex. for daytime recordings: 70-75% of data present, 10 of 16 hours (63%) data present. There are not set rules or standards. As this study utilises 22 hours recording (2 hours permitted for charging), the study team decided on the following limits: 70% for the day and 60% for the night. The % is set lower for the night as it was recognised that subjects may have more problems with night (either due to their disease, or with the technology) and so the amount of valid usable data for a night might be expected to be less. [Tudor-Locke, 2012]

#### **Daytime Endpoints**

Any data point associated with a 24-hour recording period (1440 minutes), or for a partial recording period, for DAY TIME with <9.1 hours of data for the day time is considered as a data quality data point deviator.

Day = 15 hours, permit 2 hours charging = 13 hours. 70% of 13 hours = 9.1 hours. Exclude data point if active day+sedentary day = <9.1 hours

#### Night time Endpoints

Any data point for a 24-hour recording period (1440 minutes), or for a partial recording period, for NIGHT TIME with <4.2 hours of data for the night time is considered as a data quality data point deviator.

Sleep = 9 hours, permit 2 hours charging = 7hours. 60% of 7 hours = 252 mins, 4.2 hours. Exclude data point if active night +sedentary night = <4.2 hours

## Night time rest endpoints

Sleep = 9 hours, permit 2 hours charging = 7hours. 60% of 7 hours = 252 mins, 4.2 hours. Exclude data point if active night +sedentary night = <4.2 hours

# Heart Rate Variability (24 hour endpoints only)

The amount of data present over a 24-hour recording period is also important for the 24 hour endpoints for HRV: mean and variance for HRV recorded using RMSSD methods (24 hours). 24-hour RMSSD HRV data with 40% or more data present will be accepted for analysis. The number of time windows that the HRV data is determined from is recorded in the dataset from McLaren. The following data quality rule will be applied:

Number of 5-minute windows (number of data points) in 24 hrs = 288. Allow for 2 hours charging = 24. Leaves 264 data points. Ruling = require 40% or more of data present for the 24-hour time period, otherwise it is not considered as representative of 24 hours. 40% of 264 = 105.6. Therefore, exclude data point if number of 5-minute window (number of data point) < 105.

## **Speech Endpoints**

There is no data quality rule for Speech data as there are no data quality deviators, and all available data will be included in the summary and statistical analysis.

The data quality deviator flags will be populated in the data and the summary tables and figures will be produced for data with the deviator and without the data quality deviator.

Table 3 provides an overview of the planned efficacy analyses, with further details of data displays being presented in Appendix 11: List of Data Displays.

Table 3 Overview of Planned Exploratory Analyses

| Endpoint / Parameter/ | | | Α | bsolu | te | | Cha | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Display Type | Stats Analysis Summary | | | | | Individu | | | ts Ana | | | Summary | | ividu |
| | | | • | | | al | | | | | | | | al |
| | Τ | F | L | T | F[1] | F | L | Т | F | L | Т | F[1] | F | L |
| Actigraphy - feasibility | & We | ar tim | e Mea | | | | \ <u>/</u> | Ι | | | | 1 | | |
| Wear Time (active + | | | | Υ | | | Υ | | | | | | | |
| sedentary time) Duration of day time | | | | Υ | | | Υ | | | | | | | |
| wear time | | | | I | | | I | | | | | | | |
| Duration of night time | | | | Υ | | | Υ | | | | | | | |
| wear time | | | | | | | · | | | | | | | |
| Actigraphy Diary Data | - feas | ibility | meas | ures | l | | | ı | | | | • | | |
| Actigraphy Diary data) | | | | Υ | | | Υ | | | | | | | |
| (Items 2, 3, 5, 6, 8) | | | | | | | | | | | | | | |
| And Feasibility | | | | | | | | | | | | | | |
| Device impact Data – fo | easibi | lity me | easur | | ı | | | ı | | | | 1 | | |
| Device Impact | | | | Y | 41.14 | L | Υ | | · · | | | <u> </u> | | |
| Actigraphy - Day/Night | meas | ures ( | of phy | sical | activity | - exp | olorat | ory e | Hicac | y meas | sures | | | |
| 2 measures for 24-hour<br>Time Spent Active | reco | aing | perio | u: 10ta | ai ACTIVI | ty S | core a | ana IV | iaximi | ım SC | ore | | | |
| Time Spent Active | | | | | | | 1 | | | | | | | |
| Non-normalised | | | | Υ | Υ | | Υ | | | | Υ | Υ | | |
| (Average day time | | | | | • | | · | | | | • | | | |
| active and average | | | | | | | | | | | | | | |
| night time active) & | | | | | | | | | | | | | | |
| normalised | | | | | | | | | | | | | | |
| (% daytime active; % | | | | | | | | | | | | | | |
| night time active) | | | | | | | | | | | | | | |
| Over All Time Spent | | | | | | | Υ | | | | | | | |
| sedentary not lying | | | | | | | | | | | | | | |
| Non-normalised | | | | Υ | Υ | | Υ | | | | Υ | Υ | | |
| (Average day/night | | | | ' | ' | | ' | | | | ' | ' | | |
| time spent sedentary | | | | | | | | | | | | | | |
| not lying) & normalised | | | | | | | | | | | | | | |
| (% daytime sedentary | | | | | | | | | | | | | | |
| not lying; % night time | | | | | | | | | | | | | | |
| sedentary not lying) | | | | | | | | | | | | | | |
| Over All Time Spent | | | | | | | Υ | | | | · <u> </u> | | | |
| Lying | | | | | | | | | | | | | | |
| Non-normalised | | | | Υ | Υ | | Υ | | | | Υ | Υ | | |
| (Average day/night | | | | ı | l i | | I | | | | ſ | ' | | |
| over all time spent | | | | | | | | | | | | | | |
| lying) & normalised | | | | | | | | | | | | | | |
| (% daytime lying; % | | | | | | | | | | | | | | |
| night time lying) | | | | | | | | | | | | | | |
| Over All Time Spent | | | | | | | Υ | | | | | | | |
| Sedentary | | | | | | | | | | | | | | |

| Endpoint / Parameter/ | Absolute | | | | | | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Display Type | Stats Analysis Summary | | | Ind | dividu Stats Analysis | | | | nmary | Ind | lividu | | | |
| . , , , | | | | | al | | | | | • | | al | | |
| | Т | F | L | Τ | F[1] | F | L | Т | F | L | Т | F[1] | F | L |
| Non-normalised | | | | Υ | Y | | Υ | | | | Υ | Y | | |
| (Average day/night | | | | | | | | | | | | | | |
| over all time spent | | | | | | | | | | | | | | |
| sedentary) & | | | | | | | | | | | | | | |
| normalised | | | | | | | | | | | | | | |
| (% daytime sedentary; | | | | | | | | | | | | | | |
| % night time | | | | | | | | | | | | | | |
| sedentary) | | | | | | | | | | | | | | |
| Total Activity Score | | | | Υ | Υ | | Υ | | | | Υ | Υ | | |
| Day/Night | | | | | | | | | | | | | | |
| (Total Day time | | | | | | | | | | | | | | |
| Activity score/hour; | | | | | | | | | | | | | | |
| Total Night Time | | | | | | | | | | | | | | |
| Activity score/hour) | | | | | | | | | | | | | | |
| Total Activity Score – | | | | Υ | Υ | | Υ | | | | Υ | Υ | | |
| 24 hour | | | | | | | | | | | | | | |
| (derived by adding up | | | | | | | | | | | | | | |
| the day & night scores) | | | | | | | | | | | | | | |
| Maximum Score –24 | | | | Υ | Υ | | Υ | | | | Υ | Υ | | |
| Hour | | | | | | | | | | | | | | |
| (Maximum score of | | | | | | | | | | | | | | |
| day OR night for each | | | | | | | | | | | | | | |
| 24-hour recording) | | | | | | | | | | | | | | |
| And Average of 3 | | | | | | | | | | | | | | |
| values | | | | | | | | | | | | | | |
| Active Periods | | | | Υ | Υ | | Υ | | | | | | | |
| (Numbers) | | | | | | | | | | | | | | |
| normalised / hr | | | | | | | | | | | | | | |
| Active Periods | | | | Υ | Υ | | Υ | | | | Υ | Υ | | |
| (Duration) | | | | | | | | | | | | | | |
| Relationship between | Υ | Υ | | | | | | Υ | Υ | | | | | |
| the ALSFRS and | | | | | | | | | | | | | | |
| actigraphy measures | | | | | | | | | | | | | | |
| <b>Actigraphy - Night Tim</b> | e Resi | t Endp | oints | - exp | loratory | effic | cacy r | neas | ures | | | | | |
| Number Night Time | | | | Υ | Υ | | Υ | | | | Υ | Υ | | |
| Movement | | | | | | | | | | | | | | |
| Episodes/Hr | | | | | | | | | | | | | | |
| (use average) | | | | | | | | | | | | | | |
| Percent Time Night- | | | | Υ | Υ | | Υ | | | | Υ | Υ | | |
| time Rest Efficiency | | | | | | | | | | | | | | |
| (use average) | | | | | | | | | | | | | | |
| Rest Fragmentation | | | | Υ | Υ | | Υ | | | | Υ | Υ | | |
| Index | | | | | | | | | | | | | | |
| (use average) | | | | | | | | | | | | | | |
| Average Duration | | İ | | Υ | Υ | | Υ | | | | Υ | Υ | | |
| Movement Episodes | | | | | | | | | | | | | | |

| Endpoint / Parameter/ | Absolute | | | | | | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Display Type | Stat | s Ana | s Analysis | | nmary | | ividu<br>al | | its Ana | | | nmary | | ividu<br>al |
| | Т | F | L | Т | F[1] | F | L | Τ | F | L | Т | F[1] | F | L |
| <b>Data Quality Deviators</b> | | | | | | | | | | | | | | |
| Data Quality Deviators for Actigraphy | | | | Y | | | | | | | | | | |
| Data Quality Deviators<br>for Heart Rate<br>Variability | | | | Y | | | | | | | | | | |
| Reconciliation for Action | graph | y and | Diary | Data | | | | • | • | • | • | • | | |
| Reconciliation of<br>Actigraphy and Diary<br>Data | | | | Y | | | | | | | | | | |
| <b>Heart Rate Variability M</b> | leasu | res (n | nean 8 | & varia | nce) - e | xplo | rator | y effic | cacy n | neasu | res | | | |
| LF/HF Lying | | | | Υ | Υ | | Υ | | | | Υ | Υ | | |
| LF/HF Active | | | | Υ | Υ | | Υ | | | | Υ | Υ | | |
| LF/HF Sedentary not lying | | | | Y | Υ | | Υ | | | | Υ | Υ | | |
| LF/HF Active Minus<br>Lying | | | | Y | Y | | Υ | | | | Υ | Υ | | |
| LF/HF Sedentary not lying minus Lying | | | | Y | Y | | Υ | | | | Υ | Υ | | |
| RMSSD (24 hr average) | | | | Y | Y | | Υ | | | | Υ | Y | | |
| Relationship between<br>the ALSFRS and<br>biotelemetry measures<br>of HRV. | Y | Y | | | | | | Y | Y | | | | | |
| Quantitative Speech Te | etina | - evnl | orato | ry effic | acy me | asıır | 20 | | | | | | | |
| Change over time in digital speech measures (Group by test) (Test details are in Section 9.4.3) | | | | Y | Y | | Y | | | | Y | Y | | |
| Relationship between<br>the ALSFRS and<br>digital measures of<br>speech. | Y | Y | | | | | | Y | Y | | | | | |
| Relationship between Forced Vital Capacity (FVC) and digital measures of speech. | Y | Y | | | | | | Y | Y | | | | | |
| ALSFRS-R | | | | | | | | | | | | | | |
| ALSFRS-R Total Score | | | | Υ | Υ | | Υ | | | | Υ | Υ | | |
| FVC | | | | | | | | | | | | | | |
| FVC | | | | Υ | Υ | | Υ | | | | Υ | Υ | | |

# NOTES:

[1] The figures are plotted using the absolute values over time and relative rate of decline of related endpoints. See

Section 7.1.2 for details.

- T = Table, F = Figure, L =Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

# 7.1.2. Planned Statistical Exploratory Analyses

#### **Statistical Analyses**

#### Endpoint(s)

- Movement/physical activity (Actigraphy) endpoints as measured by the accelerometer device.
   See Section 2.2 for details.
- Heart rate variability endpoints as measured by the electrode device. See Section 2.2 for details.
- Speech endpoints. See Section 2.2 for details.
- ALSFRS-R total score and ALSFRS-R scores for 4 domains: gross motor activity, fine motor activity, bulbar and respiratory function
- FVC

# **Model Specification**

## Descriptive Statistics

- Actigraphy
  - The absolute, change from baseline, and the relative rate of decline for Actigraphy related endpoints will be summarized for each protocol time point using the FAS population
  - The monthly rate of decline for the whole study period for Actigraphy related endpoints will be summarized using the FAS population
  - The absolute values over time and relative rate of decline of Actigraphy related endpoints along with the total score over time and relative rate of decline of ALSFRS-R will be plotted against time (X), respectively.
- Heart Rate Variability
  - The absolute values, change from baseline, and the relative rate of decline for HRV related endpoints (Mean & Variance for the LF/HF and 24 hours RMSSD analyses) will be summarized for each protocol time point using the FAS population
  - The monthly rate of decline for the whole study period for HRV related endpoints (Mean & Variance for the LF/HF and 24 hours RMSSD analyses) will be summarized using the FAS population
  - The absolute values and relative rate of decline of HRV related endpoints (Mean & Variance for the LF/HF and 24 hours RMSSD analyses) along with the absolute and relative rate of decline of ALSFRS-R will be plotted against time (X) respectively.
  - The Average Value and the raw data of the endpoints from McLaren will be listed

#### Speech assessment

## **Statistical Analyses**

- The absolute values, change from baseline, and the relative rate of decline for Speech related endpoints will be summarized for each protocol time point using the FAS population
- The monthly rate of decline for the whole study period for Speech related endpoints will be summarized using the FAS population
- The absolute values and relative rate of decline of Speech related endpoints along with the absolute values and relative rate of decline of ALSFRS-R total score and FVC values will be plotted against time (X), respectively.

#### • Correlation Analysis

An estimate of the between-subject correlation and the within-subject correlation will be obtained using the method described in Roy, 2006. The between-subject correlation will characterize whether subjects with greater decrease in the endpoint also tend to have the greater change in ALSFRS-R. The within-subject correlation will describe whether a decrease in one endpoint within an individual is associated with a decrease in the other endpoint.

A mixed effect model with the change from baseline in the endpoints and the change from baseline in the ALSFRS-R score as dependent variables will be fitted. An indicator variable to distinguish the two endpoints will be fitted as a fixed effect and a random effect. Other explanatory covariates will be fitted as fixed effects, as appropriate.

The RANDOM and REPEATED statements will be used to specify the structure of the covariance matrix for the two responses. The RANDOM statement will be used to specify an unstructured variance-covariance structure for the two responses. The REPEATED statement will be used to specify the variance covariance matrix for the error terms in the model. The structure of the variance covariance matrix is constructed by taking the Kronecker product of an unstructured matrix, which models the covariance for the two endpoints, with an unstructured or autoregressive (AR (1)) covariance matrix which models the covariance for the 2 repeated measures across visits.

If the data is not sufficient to allow for convergence of the model, then alternative variance covariance matrices may be considered. If convergence of the model parameters still cannot be achieved, the approach by Bland, 1995 will be used to estimate the within subject correlation.

# Actigraphy

- The absolute values and change from baseline for the actigraphy endpoints will be analyzed for correlation with absolute values and change from baseline of Total score of ALSFRS-R, respectively.
- The absolute values and change from baseline in the time spent active (day only), Time Spent sedentary not lying (day only), Time Spent Lying (day only), Time Spent Sedentary (day only), Total Activity Score (By 24 Hour and by Day), Maximum Score(By 24 Hour and by Day), Active Periods (Numbers) (day only), Active Periods (Duration) (day only) will be analysed for correlation with the absolute values and change from

## **Statistical Analyses**

baseline to the-gross motor domain and fine motor domain of ALSFRS-R, respectively.

 For the above endpoints analyzed for correlation, scatter plots will be done

The correlation analysis will be performed on both non normalized and normalized data.

Only the quality data (i.e. the data without the data quality deviators as defined in Section 7.1.1) will be used for the statistical analysis.

#### Heart Rate Variability

- The absolute values and change from baseline in the heart rate variability endpoints will be analyzed for correlation with the absolute values and change from baseline in the Total score of ALSFRS-R, respectively.
- For the above endpoints analyzed for correlation, scatter plots will be done

Only the quality data will be used for the statistical analysis.

#### Speech assessment

- The absolute values and change from baseline in the speech endpoints will be analyzed for correlation with the absolute values and change from baseline in the Total ALSFRS-R, respectively.
- The absolute values and change from baseline in the speech endpoints will be analyzed for correlation with the absolute values and change from baseline of bulbar domain and respiratory domain of ALSFRS-R, respectively.
- The absolute values and change from baseline in the speech endpoints will be analyzed for correlation with the absolute values and change from baseline in the FVC, respectively.

Only the quality data will be used for the statistical analysis.

# **Model Results Presentation**

#### Descriptive Statistics

- Data listings
- Summary tables
- Visualization graphs

#### Correlation Analysis

- Result tables
- Visualization graphs

# 7.2. Safety Analyses

# 7.2.1. Overview of Planned Analyses

The safety analyses will be based on the "Safety" population, unless otherwise specified.

Table 4 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 11: List of Data Displays.

Table 4 Overview of Planned Safety Analyses

| Endpoint / Parameter/ Display Type | Absolute | | |
|---|---|---|---|
| | Sun | nmary | Individual |
| | T | F | L |
| Adverse Events (AEs) | | | |
| All AEs by SOC | Υ | | Υ |
| Serious AEs by SOC | Υ | | Υ |
| AEs Leading to Withdrawal from Study by SOC and PT | Υ | | Υ |
| AEs based on Intensity | Υ | | Υ |
| Relationship Between AE SOCs, PT & Verbatim Text | | | Υ |
| Death | | | |
| Number of deaths | Υ | | Υ |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, SOC = System Organ Class, PT = Preferred Term.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

# 8. REFERENCES

Bland JM, Altman DG. Calculating correlation coefficients with repeated observations: Part 1—Correlation within subjects. BMJ, 1995;310:446.

Cedarbaum JM, Stambler N, Malta E, Fuller C, Hilt D, Thurmond B, Nakanishi A. The ALSFRS-R: a revised ALS functional rating scale that incorporates assessments of respiratory function. BDNF ALS Study Group (Phase III), J Neurol Sci. 1999 Oct31;169(1-2):13-21.

Clavelou P, Blanquet M, Peyrol F, Ouchchane L, Gerbaud L. Rates of progression of weight and forced vital capacity as relevant measurement to adapt Amyotrophic Lateral Sclerosi management for patient – Result of a French multicentre cohort survey. Journal of the Neurological Sciences. 2013; 331:126-131.

Cudkowicz M, Qureshi M, Shefner J. Measures and Markers in Amyotrophic Lateral Sclerosis. The Journal of the American Society for Experimental NeuroTherapeutics. 2004;1:273-283.

Czaplinski A, Yen AA, Appel SH. Forced vital capacity as an indicator of survival and disease progression in an ALS clinic population. J Neurol Neurosurg Psychiatry. 2006;77:390-392.

GlaxoSmithKline Document Number 2014N211002\_02 Study ID MID201283. An Exploratory Study to Investigate the Use of Biotelemetry to Identify Markers of Disease Progression in Subjects with Amyotrophic Lateral Sclerosis. Effective date 21-SEP-2015 (Study Protocol)

Roy A. Estimating Correlation Coefficient between Two Variables with Repeated Observations using Mixed Effects Model. Biometrical Journal. 2006; 48(2), 286–301

Tudor-Locke C, Camhi SM, Troiano RP. A Catalog of Rules, Variables, and Definitions Applied to Accelerometer Data in the National Health and Nutrition Examination Survey, 2003–2006. Prev Chronic Dis 2012;9:110332.

# 9. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 9.1 | Appendix 1: Time and Events |
| Section 9.2 | Appendix 2: Treatment States & Phases |
| Section 9.3 | Appendix 3: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 9.4 | Appendix 4: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Efficacy |
| Section 9.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 9.6 | Appendix 6: Multicentre Studies |
| Section 9.7 | Appendix 7: Examination of Covariates and Subgroups |
| Section 9.8 | Appendix 8: Multiple Comparisons and Multiplicity |
| Section 9.9 | Appendix 9: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | endices |
| Section 9.10 | Appendix 10: Abbreviations & Trade Marks |
| Section 9.11 | Appendix 11: List of Data Displays |

#### 9.1. **Appendix 1: Time & Events**

#### 9.1.1. **Protocol Defined Time & Events**

Table 1 Time and Events - Pilot Phase

| Procedures | Clinic Visit | Home<br>Monitoring | Telephone<br>Contact <sup>a</sup> | Repeat | Home<br>Monitoring <sup>b</sup> | Telephone | 200 M200 |
|---|---|---|---|---|---|---|---|
| | Screening<br>Day 0 | (~ 3 days) | (TC) | Clinic Visit <sup>b</sup> | (~ 3 days) | Contact <sup>a,b</sup> | EWD |
| Informed consent | X | 1 | | | i i | | |
| Eligibility criteria | X | | | | İ | i i | |
| Demography | X | | | | | | |
| Medical and ALS history | X | i i | | | | | |
| Brief neurological exam | Х | 1 | | Х | * | | |
| AEs/SAEs | X | | X | Χ | | Χ | Χ |
| Sensor placement | X | Χ | | Х | χ | | |
| Reference tasks | X | | | Χ | | | |
| Subject completes diary | | Χ | | | Χ | | |
| Site obtains diary information | | | Χ | | | Х | Χ |
| Device impact questionnaire | | | X | | | Χ | Χ |

a. Telephone contact to follow the 3-day home monitoring period to ensure the subject has completed the home monitoring period, diary, and to assess AEs, as appropriate. The expectation is that this call would occur on the first weekday following the home monitoring period.

Table 2 Time and Events - Core Study Phase

| | Screen/Baseline<br>Day 1/Week 0 | Weeks<br>0, 4, 8 | Week<br>12 | Weeks<br>12, 16, 20 | Week 24 | Weeks<br>24, 28, 32 | Week 36 | Weeks<br>36, 40, 44, 48° | Week 48 or<br>EWD |
|---|---|---|---|---|---|---|---|---|---|
| Study Day/Week <sup>a</sup> | Clinic<br>Visit 1 <sup>b</sup> | Home<br>Monitoring<br>(~3 days) | Clinic<br>Visit 2 | Home<br>Monitoring<br>(~3 days) | Clinic Visit | Home<br>Monitoring<br>(~3 days) | Clinic<br>Visit 4 | Home<br>Monitoring<br>(~3 days) | Clinic Visit 5 |
| Procedures | - 45 | | | · | 65 | tir 30 - 70000<br>Yu | C 10 | 7.18 S.C.116. 11 | |
| Informed consent | ΧÞ | | | | | | | | |
| Eligibility criteria | Χp | | | | | | | | |
| Demography | Χp | | | | | | | | |
| Medical and ALS history | ΧÞ | | | | | | | | |
| Neurological exam | X | | | | | | j j | | |
| Smoking details | X | | Х | | Χ | | Χ | | X |
| Brief neurological exam | 8 | | X | | Х | | Χ | | X |
| AEs/SAEs <sup>d</sup> | X | X | Х | X | Χ | X | Χ | Χ | Х |
| Concomitant medicationse | X | X | Х | X | Х | X | Χ | Χ | Х |
| ALSFRS-Re | X | X | Χ | X | Χ | Χ | Χ | X | X |
| FVC | X | | X | | X | | X | | X |
| Speech assessment | X | | X | | X | | Χ | | X |
| Sensor placement | X | X | X | X | X | Χ | Χ | Х | X |
| Reference tasks | X | | X | | X | | Χ | | X |
| Device impact questionnaire | | | Х | 3 | X | | Χ | | X |
| Subject completes diary | | X | | X | | X | | X | |
| Site obtains diary information <sup>f</sup> | | Х | Х | Х | Х | X | Χ | Χ | Х |
| Follow-up Telephone Contact9 | | X | | X | | Χ | * | Χ | |

Clinic visits and home monitoring periods should be conducted within ±7 days of the scheduled visit/home period and should be scheduled according to the Baseline Visit.
 Subjects transitioning from the Pilot Phase do not need to perform these procedures.

b. May be repeated as necessary

c. The Week 48 home monitoring period will occur the three days prior to the Week 48 in-clinic visit (Visit 5).

Assessed in clinic at Weeks 0, 12, 24, 36, and 48 and by telephone at Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44.

E. Assessed in clinic at Weeks 0, 12, 24, 36, and 48 and by telephone at Weeks 4, 8, 16, 20, 28, 32, 40, and 44.

Diary information should be obtained by telephone at Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44.

g. Telephone contact to follow each 3-day home monitoring period. The expectation is that this call would occur on the first weekday following the home monitoring period.

# 9.2. Appendix 2: Study States and Phases

# 9.2.1. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Onset Time Since<br>1st (Days) | If Start Date of wearing the device of date of first protocol specified procedure > AE Onset Date = AE Onset Date - Start Date of wearing the device If Start Date of wearing the device or date of first protocol specified procedure ≤ AE Onset Date = AE Onset Date - Start Date of wearing the device +1 Missing otherwise. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Study-related | If relationship to study participation marked 'YES' on [Inform/CRF OR value is missing]. |

Note: wearing the device refers to either the at home monitoring, or the use of the device to carry out the in clinic set reference tasks.

# 9.3. Appendix 3: Data Display Standards & Handling Conventions

## 9.3.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | |
|---|---|
| | Data Displays for Reporting |
| Code | Description |
| Α | Mega Faros Device + Fast fix |

#### 9.3.2. Baseline Definition & Derivations

#### 9.3.2.1. Baseline Definitions

For all endpoints the baseline value will be the latest assessment prior to or at the baseline visit (Visitnum=10 or 90), with the following exceptions which may use the TC at week 0 (Visitnum=100) if available:

- Actigraphy endpoints
- HRV endpoints
- Speech endpoints
- o ALSFRS-R
- o FVC

For all endpoints this will be referred to as Baseline, Week 0.

#### 9.3.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Baseline Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Baseline Visit Value – Baseline) / Baseline] |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 9.3.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.

# 9.3.3. Reporting Process & Standards

| Reporting Process | |
|---|---|
| Software | |
| The currently support of the currently su | pported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server | :UK1salx00175 |
| HARP Area | :175\gsk1223249\mid201283 |
| QC Spreadsheet | : Mc Laren-QC Sheet |

#### **Reporting Process**

## **Analysis Datasets**

Analysis datasets will be created according to IDSL standards.

#### **Generation of RTF Files**

• RTF files will be generated for all the summary tables.

# **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - o 4.03 to 4.23: General Principles
  - o 5.01 to 5.08: Principles Related to Data Listings
  - o 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables.
  - If unscheduled visits are included, provide details of how summaries will be displayed (i.e. unscheduled visits will be slotted to closest planned visit).
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

#### **Descriptive Summary Statistics**

| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
|--------------------|--------------------------------------------|
| Categorical Data | N, n, frequency, % |
| Cranbical Biombora | |

#### **Graphical Displays**

Refer to IDSL Statistical Principals 7.01 to 7.13.

# 9.4. Appendix 4: Derived and Transformed Data

#### **9.4.1.** General

#### **Multiple Measurements at One Time Point**

 For the ALSFRS-R, if the closest assessment is not evaluable, the other assessment would be used.

# **Study Day**

- Calculated as the number of days from baseline visit (visitnum=10 or 90)
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Baseline Visit Date → Study Day = Ref Date Baseline Visit Date
  - Ref Data ≥ Baseline Visit Date → Study Day = Ref Date Baseline Visit Date + 1

# 9.4.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### **Adverse Event**

For this non-drug study, an AE is any untoward medical occurrence in a clinical investigation subject which, in the opinion of the investigator, is related to a protocol-mandated procedure or one of the devices used by the subject during the study.

# 9.4.3. Exploratory

#### **ALSFRS-R Total Score**

The ALS functional rating scale – revised (ALSFRS-R) assesses the functioning of ALS subjects across 4 domains: gross motor activity, fine motor activity, bulbar and respiratory function. The ALSFRS-R [Cedarbaum, 1999] consists of 12 questions each of which are scored on a 5-point scale from 0-4, where 4 is the best possible outcome and 0 is the worst.

The total score will be calculated by summing responses to each of the 12 individual questions. The maximum total score is therefore 48, lower scores indicate worse functioning. If there are any missing questions, then the total score will be set to missing.

ALSFRS will be grouped to four different domains: Fine motor, Gross motor, Respiratory and Bulbar Domain [Cedarbaum, 1999]

#### **FVC**

FVC is a measure of respiratory function and is the volume of air that can forcibly be blown out after a single, full breath. FVC is a sensitive measure of ALS disease progression, is used as a standard test for ALS management, and is recommended as a secondary outcome measure in ALS clinical trials [Cudkowicz, 2004; Czaplinski, 2006; Clavelou, 2013].

FVC will be performed by experienced site personnel according to local protocol using a calibrated spirometer. Every effort should be made to have the same individual perform the FVC for a given subject throughout the study. For each time point, the best FVC result (in litres) will be recorded in the eCRF.

# Relative Rate of Decline and Monthly Rate of Decline (Slope)

# Relative Rate of Decline = Value at a time point - Value at the Baseline Value at the Baseline

Monthly rate of decline at each visit

Change from baseline of the endpoint at each post-baseline visit

Study day/30.4

Monthly Rate of Decline= Average of Monthly Rate of Decline at each visit and is populated only for the last visit.

For Monthly Rate of Decline, if an assessment took place over a number of consecutive days then the average of that will be taken and the recent visit (last time point) will be considered to calculate study day.

#### Actigraphy

Activity classifiers = Active / lying / "sedentary not lying".

NMTMSG – expected to be 24 hr (1440 mins) but could be less if partial recording day NMTMSG = Active, lying, "sedentary not lying", off

Each activity classifier & activity endpoint is recorded by McLaren TWICE, once for day time once for night time.

1440 = day time Active, day time lying, day time "sedentary not lying", day time off + night time Active, night time lying, night time "sedentary not lying", night time off

Therefore, wear time = 1440 minus [day off time + night off time]

Off time here represents the time that the sensor was either switched off or the patient was not wearing it (or both).

For all the parameters, derivation will be done twice – one with all data and one with the quality data (i.e., excluding data quality deviators).

For each endpoint for the CSR (& interpretation of the study) 3 splits of data will be reported:

- Day time activity endpoints from McLaren
- Night tine activity endpoints from McLaren
- 24 hour endpoints <u>derived by GSK</u> add day time + night time values

| DED!\ (ED | lar e e e | T = |
|---|---|---|
| DERIVED | Wear time (mins) | Time Active + Time sedentary [where time sedentary = time lying + time sedentary not lying] |
| DERIVED | Duration of day time wear time (mins) | Day time wear time = day time Active + day time lying + day time "sedentary not lying" |
| DERIVED | Duration of night time wear time (mins) | Night time wear time = night<br>time Active + night time lying +<br>night time "sedentary not<br>lying" |
| ACTIVETM | Overall time spent active Average day time active | Number mins per day/night for 24-hour recording period |
| | % daytime ACTIVE % night time ACTIVE | Add up the total amount of time active across all the recording periods and divide by the number of recording periods. |
| | | 1 value per subject per time point |
| | | DAYTIME ACTIVETM (Day 1+2+3) divided by total amount of day time duration across the 3 recording days – expressed as a % |
| | | Where total amount of daytime duration = [Day 1-day time ACTIVETM + day time LIETM + day time "sedentary not lying" – SEDTMNL] + Day 2 (ditto) + Day 3 [ditto] NIGHTTIME ACTIVETM (Day |

| SEDTMNL | Overall time spent sedentary not lying % daytime SEDENTARY NOT LYING % night time SEDENTARY NOT LYING | 1+2+3) divide by total amount of night time duration across the 3 recording days – expressed as a % Where total amount of night time duration = [Day 1-night time ACTIVETM + night time LIETM + night time "sedentary not lying" – SEDTMNL] + Day 2 (ditto) + Day 3 [ditto] Needs the same approach as above |
|---|---|---|
| LIETM | Overall time spent lying % daytime LYING % night time LYING | Needs the same approach as above |
| SEDENTM | Over all time spent sedentary % daytime SEDENTARY % night time SEDENTARY | Same Approach as above |
| OFFTM | Time spent with sensor | |
| ACTIVISC | Total activity score 24- Hour Daytime total activity score Night time total activity score | Total Activity Score (add day + night) Day time total activity score (Day 1+2+3) divide by the total day time for that protocol time point. Night time total activity score Day (Day 1+2+3) divide by the total day time for that protocol time point. |
| MAXACTSC | The maximum score from a 1 min window in a 24-hour | 3 values per protocol time point or more if more days are |

| | | <del>, , </del> |
|---|---|---|
| | period | recorded for home monitoring. |
| | Daytime maximum activity score | Take the maximum over<br>the 3 days |
| | Daytime mean maximum activity score (mean of all recording periods) | Average over 3 days |
| | Night time maximum activity score | |
| | Night time mean maximum activity score (mean of all recording | |
| WKPER01, WKPER02,<br>WKPER05, WKPER15,<br>WKPER30 | Active Periods (Numbers) | To normalise 'Active Periods (Number)' to a per hour unit |
| With Little | | (Algorithm is given below) |
| WKPERDUR | Average duration of active periods greater than 1 minute. | |

# To normalise 'Active Periods (Number)':

- 1. Add up the total number of 'active periods' for the recording periods (value 1).
  - Please note this is done by adding the 'number of active periods (all the categories)1min<x<2min' + 'number of active periods 2min<x<5min' + 'number of active periods 5min<x<15min' + 'number of active periods 15min<x<30min' + 'number of active periods >30min'
- 2. Calculate the 'wear time' for the recording period in days(i.e. minutes/ 1440). (value 2).
  - Please remember that 'wear time = active + sedentary time' for the recording period (either day time or night time)
- 3. Value 1 / Value 2 is the normalised measure required

#### Rules for reconciliation of Actigraphy and Diary data

Actigraphy and Diary data will be reconciled and a frequency table on the rules below will be summarized;

Rule1: Subjects present both in Actigraphy and Diary data

Rule2: Subjects present only in Actigraphy data

Rule3: Subjects present only in Diary data

# Night Time Endpoints

These endpoints need to be reported as the "average" or "mean" for each protocol time point (due to the amount of day or night time not matching a protocol day or night)

| CODE | DESCRIPTION |
|---|---|
| COBE | BESONII HON |
| NNTMTEPHR | Number Night Time Movement Episodes/Hr |
| NTRESTEF | Percent Time Night-time Rest Efficiency |
| RFRGI | Rest Frag Index=Move Time/Num Movement Episode |
| AVGDURMTE | Average Duration Movement Episodes |
| Number Night Time Movement Episodes/Hr. NNTMTEPHR | Limitations of each 24-hour recording period = the 24-hour recording periods do NOT match protocol days, due to the mixed start times that are governed by the sensor "activation." (first data recorded by the sensor) – as such reporting the data out by recording day does NOT make sense, the data must be reported over the 3 days for each protocol timepoint (ie data need to be averaged out). A note pertaining to this must be added to any data that lists out the raw data for each recording period. |
| | Average number night time movements/hour (Day 1+2+3) divide by 3, ie Day 1 + Day 2 etc. / actual number of recording periods at each time point (sometimes there are more or less values at each protocol time point) |
| Percent Time Night-time Rest Efficiency NTRESTEF | Core study phase only. Limitations as above |
| | Average % time night time rest efficiency (Day 1+2+3 values) divide by 3, ie Day 1 value + Day 2 value etc. / actual number of recording periods at each time point (sometimes there are more or less values at each protocol time point) |
| Rest Frag Ind=Move Time/Num RFRGI Movement Episode | Core study phase only. Limitations as above |
| N Not iviovement Episode | Average night time rest fragmentation index (Day 1+2+3 values) divide by 3, ie Day 1 value + Day 2 value etc. / actual number of recording periods at each time point (sometimes there are more or less values at each protocol time point) |

| Avg Duration Movement Episodes AVGDURMTE | Done for each 24 hours' period But again, need 1 value for protocol time point. An average of the average over 3 days. – Use the number of active periods in the categories above – add up to derive a total, use |
|---|---|
| | that total to create a more accurate average. Average duration of movement disorders = values [Day 1 + day 2 + day 3]/total number of night time movements [Days 1+2+3] |

# **Speech Assessments**

The 4 tests for speech assessments are:

- Short ah
  - o Central tendency of fundamental F0, relative jitter, relative shimmer
- Long ah
  - o Central tendency of fundamental F0, relative jitter, relative shimmer
- Single word doily
  - O Average phoneme rate, average phonation time
- Running speech (bamboo passage)
  - o Speaking rate % pause time

| CODE | DESCRIPTION |
|---|---|
| AA001 | Central tendency of fundamental F0 |
| | (code 001: short ah) |
| HZ | (code 002: long ah) ?? middle five seconds of the phonation interval?? |
| AA002 | Relative Jitter |
| | (code 001: short ah) |
| % | (code 002: long ah) |
| AA003 | Relative Shimmer |
| | (code 001: short ah) |

| % | (code 002: long ah) |
|---|---|
| AA004<br>(Hz/s) | Average phoneme rate (Phoneme – subpart of word) code 003: "single word" doily |
| AA005 | Average phonation time |
| (s) | code 003: "single word" doily |
| AA007 | % pause time |
| % | (Code 004: running speech) |
| AA008 | Speaking rate |
| (WPM) | (Code 004: running speech) |

# Heart Rate Variability (all LF/HF HRV metrics are over 5 minutes' windows)

HRV data are captured for each of the activity classifiers: Active + Lying + "sedentary not lying". "Lying minus active" and "Lying minus sedentary not lying" is derived based on the following:

| MLFHFN | Mean LF/HF (Avg over 5 min windows of lying down) | Use the sum of the means over each recording day (Day 1 + Day 2 + Day 3) divided by the total number of recording points over the 3 days (number Day 1+2+3) (number of lying periods of good enough quality to obtain HRV from) |
|---|---|---|
| VLFHFN | Var of LF/HF (Avg over 5 min windows of lying down) | Use the sum of the variances over each recording day (Day 1 + Day 2 + Day 3) divided by the total number of recording points over the 3 days (number Day 1+2+3) (number of lying periods of good |

| Stationary = sedentary not lying | | | enough quality to obtain HRV from) |
|---|---|---|---|
| Stationary = sedentary not lying Stationary = sedentary not lying VLFHFSD Var of LF/HF (avg-stationaryday) Var of LF/HF (avg-stationaryday) Stationary = sedentary not lying period good enough quality to obtain HRV from) Stationary = sedentary not lying Was the sum of the variance over each recording day divided by the total number or sedentary not lying' period good enough quality to obtain HRV from) MLFHFAD Mean LF/HF (avg-daytime activity) Mean LF/HF (avg-daytime activity) Var of LF/HF (avg-daytime activity) Var of LF/HF (avg-daytime activity) Var of LF/HF (avg-daytime activity) Use the sum of the means over each recording day divided by the total number or active periods of good enouguality to obtain HRV from) Derive 1 average value for each protocol time point, Use the sum of the variance over each recording day divided by the total number or each protocol time point, Use the sum of the variance over each recording day divided by the total number recording points (number or each protocol time point, over each recording day divided by the total number or each protocol time point, over each recording day divided by the total number or each protocol time points (number or each protocol time point). | MLFHFSD | ` ` ` | Derive 1 average value for each protocol time point, |
| VEFHFSD Var of LF/HF (avg-stationary-day) Var of LF/HF (avg-daytime activity) Var of LF/HF (avg-daytime activity) Var of LF/HF (avg-daytime activity) Perive 1 average value for each protocol time point, Use the sum of the variance over each recording day divided by the total number or 'sedentary not lying' periods good enough quality to obtat HRV from) MEFHFAD Mean LF/HF (avg-daytime activity) Derive 1 average value for each protocol time point, Use the sum of the means over each recording day divided by the total number recording points (number or active periods of good enouguality to obtain HRV from) VLFHFAD Var of LF/HF (avg-daytime activity) Derive 1 average value for each protocol time point, Use the sum of the variance over each recording day divided by the total number recording points (number or active periods of good enouguality to obtain the variance over each recording day divided by the total number recording points (number or active periods of good enouguality to obtain the variance over each recording day divided by the total number recording points (number or active periods of good enouguality to obtain the variance over each recording day divided by the total number recording points (number or active periods of good enough quality to obtain the variance over each recording day divided by the total number or active periods of good enough quality to obtain the variance over each recording day divided by the total number recording points (number or active periods of good enough quality to obtain the variance over each recording day divided by the total number or active periods of good enough quality to obtain the variance over each recording day divided by the total number or active periods of good enough quality to obtain the variance over each recording day divided by the total number or active periods of good enough quality to obtain the variance over each recording day divided by the total number or active periods of good enough quality to obtain the variance over each recording d | | , , | over each recording day (Day 1 + Day 2 + Day 3) divided by the total number of recording points over the 3 days (number Day 1+2+3) (number of 'sedentary not lying' periods of good enough quality to |
| Stationary = sedentary not lying Stationary = sedentary not lying MLFHFAD Mean LF/HF (avg-daytime activity) MLFHFAD Mean LF/HF (avg-daytime activity) Mean LF/HF (avg-daytime activity) Derive 1 average value for each protocol time point, Use the sum of the means over each recording day divided by the total number recording points (number or active periods of good enouguality to obtain HRV from) VLFHFAD Var of LF/HF (avg-daytime activity) Derive 1 average value for each protocol time point, Use the sum of the variance over each recording day divided by the total number recording points (number or each protocol time point, Use the sum of the variance over each recording day divided by the total number recording points (number or active periods of good enough divided by the total number or active periods o | VLFHFSD | ` • | Derive 1 average value for |
| activity) each protocol time point, Use the sum of the means over each recording day divided by the total number recording points (number or active periods of good enouguality to obtain HRV from) VLFHFAD Var of LF/HF (avg-daytime activity) Derive 1 average value for each protocol time point, Use the sum of the variance over each recording day divided by the total number recording points (number or active periods of good enougeness) | | , , | divided by the total number of recording points (number of 'sedentary not lying' periods of good enough quality to obtain |
| over each recording day divided by the total number recording points (number of active periods of good enouguality to obtain HRV from) VLFHFAD Var of LF/HF (avg-daytime activity) Derive 1 average value for each protocol time point, Use the sum of the variance over each recording day divided by the total number recording points (number of active periods of good enougeness) | MLFHFAD | ` ` ` ` | Derive 1 average value for each protocol time point, |
| VLFHFAD Var of LF/HF (avg-daytime activity) Derive 1 average value for each protocol time point, Use the sum of the variance over each recording day divided by the total number recording points (number of active periods of good enough) | | | over each recording day<br>divided by the total number of<br>recording points (number of<br>active periods of good enough |
| over each recording day divided by the total number or active periods of good enough | VLFHFAD | , , | Derive 1 average value for |
| | | | Use the sum of the variances over each recording day divided by the total number of recording points (number of active periods of good enough quality to obtain HRV from) |
| MRMSSD Mean RMSSD (24 hr avg) VRMSSD Var of RMSSD (24 hrs avg) | | \ | |

- HRV effect of being upright = LF/HF stationary minus LF/HF lying
- HRV effect of activity = LF/HF active (MLFHFAD) minus LF/HF lying (MLFHFN)
# 9.5. Appendix 5: Premature Withdrawals & Handling of Missing Data

### 9.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as a subject is one who has completed the study through the Week 48 visit.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

### 9.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing<br/>displays. Unless all data for a specific visit are missing in which case the<br/>data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to<br/>be missing data and should be displayed as such.</li> </ul> |
| Statistical analyses | For all other endpoints no imputation will be made for missing data. |

### 9.5.2.1. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications | The recorded partial date will be displayed in listings. |
| Adverse<br>Events | <ul> <li>Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if these results in a date prior to Day 1 and the event could possibly have occurred during the On-Device phase from the partial information, then the Day 1 date will be assumed to be the start date.</li> <li>The AE will then be considered to start on-device (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |

## 9.6. Appendix 6: Multicentre Studies

This study aims to enrol subjects using two sites based in the UK. In this multicentre study, listings will be presented by investigative site.

## 9.7. Appendix 7: Examination of Covariates, Subgroups & Other Strata

### 9.7.1. Handling of Covariates, Subgroups & Other Strata

There was no randomisation and therefore no strata used in this study.

Due to the small number of subjects in the study, no subgroups will be specified here although subgroup analyses may take place ad hoc.

The following is a list of covariates that may be used in descriptive summaries and/ or statistical analyses (See Section 7.1.1 and Section 7.1.2 for further details).

Additional covariates of clinical interest may also be considered.

These analyses will be carried out as part of ADHOC if necessary.

| Category | Covariates and / or Subgroups |
|---|---|
| Correlation of ALSFRS-R and movement actigraphy data/ HRV data | In additional to the model described in Section 7.1.2, the following explanatory variables may be considered: Baseline value for each of the dependent variables being correlated Phenotype at onset: Bulbar/Limb/Other Age at baseline Sex – Male/ Female Time since onset of muscle weakness |
| Correlation of FVC/ ALSFRS-R and speech data | In additional to the model described in Section 7.1.2, the following explanatory variables may be considered: Baseline value for each of the dependent variables being correlated Phenotype at onset: Bulbar/Limb/Other Smoking status at baseline Age at baseline Sex – Male/ Female Time since onset of muscle weakness |
| Mixed model repeated measures analyses | For the MMRM Baseline, Visit, Baseline by Visit covariates will be included in model. The following explanatory variables may also be considered: • Phenotype at onset: Bulbar or Other/ Limb • Smoking status at baseline • Age at baseline • Sex – Male/ Female • Time since onset of muscle weakness |

### 9.8. Appendix 8: Multiple Comparisons & Multiplicity

As this is an exploratory study, no adjustment will be made for multiple comparisons. Assessments about the correlation between endpoints will be made on the strength of the correlation coefficients.

## 9.9. Appendix 9: Model Checking and Diagnostics for Statistical Analyses

#### 9.9.1. Statistical Analysis Assumptions

| Endpoint(s) | • | Actigraphy, HRV and Speech |
|-------------|---|----------------------------|
| Analysis | • | MMRM |

- Model assumptions will be applied, but appropriate adjustments maybe made based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.
  - In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.
  - Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.
- Distributional assumptions underlying the model used for analysis will be examined by
  obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
  values (i.e. checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

## 9.10. Appendix 10: – Abbreviations & Trade Marks

### 9.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| ALSFRS-R | Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised |
| A&R | Analysis and Reporting |
| CI | Confidence Interval |
| CS | Clinical Statistics |
| CS | Compound Symmetry |
| CSH | Heterogeneous Compound Symmetry |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| FAS | Full Analysis Set |
| FVC | Forced Vital Capacity |
| GSK | GlaxoSmithKline |
| HF | High Frequency |
| HRV | Heart Rate Variability |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| GUI | Guidance |
| LF | Low Frequency |
| MMRM | Mixed Model Repeated Measures |
| PDMP | Protocol Deviation Management Plan |
| PP | Per Protocol |
| QC | Quality Control |
| RAP | Reporting & Analysis Plan |
| RMSSD | Root Mean Square |
| SAC | Statistical Analysis Complete |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

### 9.10.2. Trademarks

| Trademarks of the GlaxoSmithKline |
|-----------------------------------|
| Group of Companies |

NONE

# Trademarks not owned by the GlaxoSmithKline Group of Companies

McLaren
Mega Faros
SAS

### 9.11. Appendix 11: List of Data Displays

### 9.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|--------------|-------------|
| Study Population | 1.1 to 1.8 | NA |
| Exploratory | 2.1 to 2.155 | 2.1 to 2.94 |
| Safety | 3.1 to 3.5 | NA |
| Section | Listi | ngs |
| ICH Listings | 1 to | 15 |
| Other Listings | 16 to | 70 |

### 9.11.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in a separate document.

| Section | Figure | Table | Listing |
|------------------|--------|---------|---------|
| Study Population | NA | NA | NA |
| Exploratory | EFF_F1 | EFF_T1 | EFF_L1 |
| Safety | NA | SAFE_T1 | SAFE_L1 |

#### NOTES:

 Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

## 9.11.3. Study Population Tables

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | |
| 1.1. | FAS | CP_ES1 | Summary of Subject Disposition | | SAC |
| 1.2. | Screen<br>Failure | ES6 | Summary of Reasons for Screen Failure | | SAC |
| 1.3. | FAS | NS1 | Summary of Number of Subjects by Country and Centre | | SAC |
| Protoco | ol Deviations | | | | |
| 1.4. | FAS | DV1 | Summary of Important Protocol Deviations | | SAC |
| Popula | tion Analysed | | | | |
| 1.5. | Enrolled | SP1 | Summary of Study Populations and Exclusions | | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.6. | FAS | DM3 | Summary of Demographic Characteristics | Add ALSFRS-R and FVC at baseline | SAC |
| 1.7. | FAS | DM5 | Summary of Race and Racial Combinations | | SAC |
| Prior ar | nd Concomitan | t Medications | | | |
| 1.8. | FAS | CM1 | Summary of Concomitant Medications | | SAC |

## 9.11.4. Exploratory Tables

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Actigra | phy - feasibility | y & Wear time Mea | asures | | |
| 2.1. | FAS | EFF_T1 | Summary of Wear Time (mins) (All data) | By visit and Overall Paginate by Pilot Phase and Core Phase | SAC |
| 2.2. | FAS | EFF_T1 | Summary of Wear Time (mins)<br>(Quality data) | By visit and Overall Paginate by Pilot Phase and Core Phase | SAC |
| 2.3. | FAS | EFF_T1 | Summary of Duration of Day Wear Time (All data) | Same as Above | SAC |
| 2.4. | FAS | EFF_T1 | Summary of Duration of Day Wear Time (Quality data) | Same as Above | SAC |
| 2.5. | FAS | EFF_T1 | Summary of Duration of Night Time Wear Time (All data) | Same as Above | SAC |
| 2.6. | FAS | EFF_T1 | Summary of Duration of Night Time Wear Time (Quality data) | Same as Above | SAC |
| _ | | | sical activity - exploratory efficacy measures | | |
| 2 meas | ures for 24-hoเ | ur recording perio | d: Total Activity Score and Maximum Score | | |
| 2.7. | FAS | EFF_T1 | Summary of Time Spent Active (All data) | Categorise into: Average Day/Night Time active %Day Time Active %Night Time Active | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.8. | FAS | EFF_T1 | Summary of Time Spent Active (Quality data) | Categorise into: Average Day/Night Time active %Day Time Active %Night Time Active | SAC |
| 2.9. | FAS | EFF_T1 | Summary of Change from Baseline of Time Spent Active (All data) | Same as Above | SAC |
| 2.10. | FAS | EFF_T1 | Summary of Change from Baseline of Time Spent Active (Quality data) | Same as Above | SAC |
| 2.11. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Time Spent Active (All data) | Same as Above | SAC |
| 2.12. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Time Spent Active (Quality data) | Same as Above | SAC |
| 2.13. | FAS | EFF_T1 | Summary of Monthly Rate of Decline of Time Spent Active (Quality data) | Same as Above | SAC |
| 2.14. | FAS | EFF_T1 | Summary of Overall Time Spent Sedentary Not Lying (All data) | Same as Above | SAC |
| 2.15. | FAS | EFF_T1 | Summary of Overall Time Spent Sedentary Not Lying (Quality data) | Same as Above | SAC |
| 2.16. | FAS | EFF_T1 | Summary of Change from Baseline of Overall Time Spent<br>Sedentary Not Lying<br>(All data) | Same as Above | SAC |
| 2.17. | FAS | EFF_T1 | Summary of Change from Baseline of Overall Time Spent<br>Sedentary Not Lying<br>(Quality data) | Same as Above | SAC |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.18. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Overall Time Spent Sedentary Not Lying (All data) | Same as Above | SAC |
| 2.19. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Overall Time Spent Sedentary Not Lying (Quality data) | Same as Above | SAC |
| 2.20. | FAS | EFF_T1 | Summary of Monthly Rate of Decline of Overall Time Spent Sedentary Not Lying (Quality data) | Same as Above | SAC |
| 2.21. | FAS | EFF_T1 | Summary of Time Spent Lying (All data) | Categorise into: Average Day/Night Overall Time Spent Lying %Day Time Lying %Night Time Lying | SAC |
| 2.22. | FAS | EFF_T1 | Summary of Time Spent Lying (Quality data) | Categorise into: Average Day/Night Overall Time Spent Lying %Day Time Lying %Night Time Lying | SAC |
| 2.23. | FAS | EFF_T1 | Summary of Change from Baseline of Time Spent Lying (All data) | Same as Above | SAC |
| 2.24. | FAS | EFF_T1 | Summary of Change from Baseline of Time Spent Lying (Quality data) | Same as Above | SAC |
| 2.25. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Time Spent Lying (All data) | Same as Above | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.26. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Time Spent Lying (Quality data) | Same as Above | SAC |
| 2.27. | FAS | EFF_T1 | Summary of Monthly Rate of Decline of Time Spent Lying (Quality data) | Same as Above | SAC |
| 2.28. | FAS | EFF_T1 | Summary of Time Spent Sedentary (All data) | Categorise into: Average Day/Night Time Spent Sedentary %Day Time Sedentary %Night Time Sedentary | SAC |
| 2.29. | FAS | EFF_T1 | Summary of Time Spent Sedentary (Quality data) | Same as Above | SAC |
| 2.30. | FAS | EFF_T1 | Summary of Change from Baseline of Time Spent Sedentary (All data) | Same as Above | SAC |
| 2.31. | FAS | EFF_T1 | Summary of Change from Baseline of Time Spent Sedentary (Quality data) | Same as Above | SAC |
| 2.32. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Time Spent Sedentary (All data) | Same as Above | SAC |
| 2.33. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Time Spent Sedentary (Quality data) | Same as Above | SAC |
| 2.34. | FAS | EFF_T1 | Summary of Monthly Rate of Decline of Time Spent Sedentary (Quality data) | Same as Above | SAC |
| 2.35. | FAS | EFF_T1 | Summary of Total Activity Score Day/Night (All data) | Categorise into: Total Day Time Activity Score Total Night Time Activity Score | SAC |

| Efficacy | r: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.36. | FAS | EFF_T1 | Summary of Total Activity Score Day/Night (Quality data) | Same as Above | SAC |
| 2.37. | FAS | EFF_T1 | Summary of Change from Baseline of Total Activity Score Day/Night (All data) | Same as Above | SAC |
| 2.38. | FAS | EFF_T1 | Summary of Change from Baseline of Total Activity Score Day/Night (Quality data) | Same as Above | SAC |
| 2.39. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Total Activity Score Day/Night (All data) | Same as Above | SAC |
| 2.40. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Total Activity Score Day/Night (Quality data) | Same as Above | SAC |
| 2.41. | FAS | EFF_T1 | Summary of Monthly Rate of Decline of Total Activity Score Day/Night (Quality data) | Same as Above | SAC |
| 2.42. | FAS | EFF_T1 | Summary of Total Activity Score – 24 Hour (All data) | | SAC |
| 2.43. | FAS | EFF_T1 | Summary of Total Activity Score – 24 Hour (Quality data) | | SAC |
| 2.44. | FAS | EFF_T1 | Summary of Change from Baseline of Total Activity Score – 24<br>Hour<br>(All data) | | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.45. | FAS | EFF_T1 | Summary of Change from Baseline of Total Activity Score – 24 Hour (Quality data) | | SAC |
| 2.46. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Total Activity Score – 24 Hour (All data) | | SAC |
| 2.47. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Total Activity Score – 24 Hour (Quality data) | | SAC |
| 2.48. | FAS | EFF_T1 | Summary of Monthly Rate of Decline of Total Activity Score – 24 Hour (Quality data) | | SAC |
| 2.49. | FAS | EFF_T1 | Summary of Maximum Score (1 min – 24 Hour Window) (All data) | Categorise into: Daytime maximum activity score Daytime mean maximum activity score (mean of all recording periods) Night time maximum activity score Night time mean maximum activity score (mean of all recording | SAC |
| 2.50. | FAS | EFF_T1 | Summary of Maximum Score (1 min – 24 Hour Window) (Quality data) | Same as above | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.51. | FAS | EFF_T1 | Summary of Change from Baseline Maximum Score (1 min – 24 Hour Window) (All data) | Same as above | SAC |
| 2.52. | FAS | EFF_T1 | Summary of Change from Baseline Maximum Score (1 min – 24 Hour Window) (Quality data) | Same as above | SAC |
| 2.53. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Maximum Score (1 min – 24 Hour Window) (All data) | Same as above | SAC |
| 2.54. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Maximum Score (1 min – 24 Hour Window) (Quality data) | Same as above | SAC |
| 2.55. | FAS | EFF_T1 | Summary of Monthly Rate of Decline of Maximum Score (1 min – 24 Hour Window) (Quality data) | Same as above | SAC |
| 2.56. | FAS | EFF_T1 | Summary of Active Periods (Numbers) (All data) | For day and night active periods separately & for each category (> 1 to <= 2 minutes, > 2 to <= 5 minutes etc. etc): Categorise into Day and Night Time Modify EFF_T1 as: Add n (%) instead of statistics Add columns for categories | SAC |
| 2.57. | FAS | EFF_T1 | Summary of Active Periods (Numbers)<br>(Quality data) | Same as Above | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.58. | FAS | EFF_T1 | Summary of Active Periods (Duration) (All data) | Categorise into Day and Night Time | SAC |
| 2.59. | FAS | EFF_T1 | Summary of Active Periods (Duration) (Quality data) | Same as Above | SAC |
| 2.60. | FAS | EFF_T1 | Summary of Change from Baseline of Active Periods (Duration) (All Data) | Same as Above | SAC |
| 2.61. | FAS | EFF_T1 | Summary of Active Change from Baseline of Periods (Duration) (Quality data) | Same as Above | SAC |
| 2.62. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Active Periods (Duration) (All data) | Same as Above | SAC |
| 2.63. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Active Periods (Duration) (Quality data) | Same as Above | SAC |
| 2.64. | FAS | EFF_T1 | Summary of Monthly Rate of Decline of Active Periods (Duration) (Quality data) | Same as Above | SAC |
| 2.65. | FAS | EFF_T3 | Statistical Analysis of Relationship between Absolute Values of Actigraphy endpoints and Absolute Value of Total ALSFRS-R | | SAC |
| 2.66. | FAS | EFF_T3 | Statistical Analysis of Relationship between Change from Baseline of Actigraphy endpoints and Change from Baseline of Total ALSFRS-R | | SAC |
| 2.67. | FAS | EFF_T3 | Statistical Analysis of Relationship between Slope of Actigraphy endpoints and Slope of Total ALSFRS-R | | SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.68. | FAS | EFF_T3 | Statistical Analysis of Relationship between Absolute Values of Actigraphy endpoints and Absolute Value of gross motor domain of ALSFRS-R | | SAC |
| 2.69. | FAS | EFF_T3 | Statistical Analysis of Relationship between Change from Baseline of Actigraphy endpoints and Change from Baseline of gross motor domain of ALSFRS-R | | SAC |
| 2.70. | FAS | EFF_T3 | Statistical Analysis of Relationship between Slope of Actigraphy endpoints and Slope of gross motor domain of ALSFRS-R | | SAC |
| 2.71. | FAS | EFF_T3 | Statistical Analysis of Relationship between Absolute Values of Actigraphy endpoints and Absolute Value of fine motor domain of ALSFRS-R | | SAC |
| 2.72. | FAS | EFF_T3 | Statistical Analysis of Relationship between Change from Baseline of Actigraphy endpoints and Change from Baseline of fine motor domain of ALSFRS-R | | SAC |
| 2.73. | FAS | EFF_T3 | Statistical Analysis of Relationship between Slope of Actigraphy endpoints and Slope of fine motor domain of ALSFRS-R | | SAC |
| Night T | ime Rest Endp | oints | | | |
| 2.74. | FAS | EFF_T1 | Summary of Number Night Time Movement (All data) | | SAC |
| 2.75. | FAS | EFF_T1 | Summary of Number Night Time Movement (Quality data) | | SAC |
| 2.76. | FAS | EFF_T1 | Summary of Change from Baseline of Number Night Time<br>Movement<br>(All data) | | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.77. | FAS | EFF_T1 | Summary of Change from Baseline of Number Night Time<br>Movement<br>(Quality data) | | SAC |
| 2.78. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Number Night Time<br>Movement<br>(All data) | | SAC |
| 2.79. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Number Night Time<br>Movement<br>(Quality Da data ta) | | SAC |
| 2.80. | FAS | EFF_T1 | Summary of Monthly Rate of Decline of Number Night Time Movement (Quality data) | | SAC |
| 2.81. | FAS | EFF_T1 | Summary of Percent Time Night-time Rest Efficiency (All data) | | SAC |
| 2.82. | FAS | EFF_T1 | Summary of Percent Time Night-time Rest Efficiency (Quality data) | | SAC |
| 2.83. | FAS | EFF_T1 | Summary of Change from Baseline of Percent Time Night-time<br>Rest Efficiency<br>(All data) | | SAC |
| 2.84. | FAS | EFF_T1 | Summary of Change from Baseline of Percent Time Night-time Rest Efficiency (Quality data) | | SAC |
| 2.85. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Percent Time Night-time Rest Efficiency (All data) | | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.86. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Percent Time Night-time Rest Efficiency (Quality data) | | SAC |
| 2.87. | FAS | EFF_T1 | Summary of Monthly Rate of Decline of Percent Time Night-time<br>Rest Efficiency<br>(Quality data) | | SAC |
| 2.88. | FAS | EFF_T1 | Summary of Rest Fragmentation Index (All data) | | SAC |
| 2.89. | FAS | EFF_T1 | Summary of Rest Fragmentation Index (Quality data) | | SAC |
| 2.90. | FAS | EFF_T1 | Summary of Change from Baseline of Rest Fragmentation Index (All data) | | SAC |
| 2.91. | FAS | EFF_T1 | Summary of Change from Baseline of Rest Fragmentation Index (Quality data) | | SAC |
| 2.92. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Rest Fragmentation Index (All data) | | SAC |
| 2.93. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Rest Fragmentation Index (Quality data) | | SAC |
| 2.94. | FAS | EFF_T1 | Summary of Monthly Rate of Decline of Rest Fragmentation Index (Quality data) | | SAC |
| 2.95. | FAS | EFF_T1 | Summary of Average Duration Movement Episodes (All data) | | SAC |
| 2.96. | FAS | EFF_T1 | Summary of Average Duration Movement Episodes (Quality data) | | SAC |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.97. | FAS | EFF_T1 | Summary of Average Change from Baseline of Duration<br>Movement Episodes<br>(All data) | | SAC |
| 2.98. | FAS | EFF_T1 | Summary of Average Change from Baseline of Duration<br>Movement Episodes<br>(Quality data) | | SAC |
| 2.99. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Duration Movement Episodes (All data) | | SAC |
| 2.100. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Duration Movement Episodes (Quality data) | | SAC |
| 2.101. | FAS | EFF_T1 | Summary of Monthly Rate of Decline of Duration Movement Episodes (Quality data) | | SAC |
| 2.102. | FAS | EFF_T3 | Statistical Analysis of Relationship between Absolute Values of Night Rest Endpoints and Absolute Value of Total ALSFRS-R | | SAC |
| 2.103. | FAS | EFF_T3 | Statistical Analysis of Relationship between Change from Baseline of Night Rest Endpoints and Change from Baseline of Total ALSFRS-R | | SAC |
| 2.104. | FAS | EFF_T3 | Statistical Analysis of Relationship between Slope of Night Rest Endpoints and Slope of Total ALSFRS-R | | SAC |

| Efficacy | r: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Heart R | ate Variability | | | | |
| 2.105. | FAS | EFF_T1 | Summary of Mean HRV LF/HF (All data) | Include: Mean HRV Lying minus active Mean HRV Lying minus 'sedentary not lying' Mean HRV Lying (average) Mean HRV Active(average) Mean HRV 'sedentary not lying' (average) | SAC |
| 2.106. | FAS | EFF_T1 | Summary of Change from Baseline of Mean HRV LF/HF (All data) | Same as above | SAC |
| 2.107. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Mean HRV LF/HF (All data) | Same as above | SAC |
| 2.108. | FAS | EFF_T1 | Summary of Monthly Rate of Decline of Mean HRV LF/HF (All data) | Same as above | SAC |
| 2.109. | FAS | EFF_T1 | Summary of Mean RMSSD (All data) | | SAC |
| 2.110. | FAS | EFF_T1 | Summary of Mean RMSSD (Quality data) | | SAC |
| 2.111. | FAS | EFF_T1 | Summary of Change from Baseline of Mean RMSSD (All data) | | SAC |
| 2.112. | FAS | EFF_T1 | Summary of Change from Baseline of Mean RMSSD (Quality data) | | SAC |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.113. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Mean RMSSD (All data) | | SAC |
| 2.114. | FAS | EFF_T1 | Summary of Relative Rate of Mean RMSSD (Quality data) | | SAC |
| 2.115. | FAS | EFF_T1 | Summary of Monthly Rate of Decline of Mean RMSSD (Quality data) | | SAC |
| 2.116. | FAS | EFF_T1 | Summary of Variance HRV LF/HF (All data) | Include: Variance HRV Lying minus active Variance HRV Lying minus 'sedentary not lying' Variance HRV Lying (average) Variance HRV Active(average) Variance HRV 'sedentary not lying' (average) | SAC |
| 2.117. | FAS | EFF_T1 | Summary of Change from Baseline of Variance HRV LF/HF (All data) | Same as above | SAC |
| 2.118. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Variance HRV LF/HF (All data) | Same as above | SAC |
| 2.119. | FAS | EFF_T1 | Summary of Monthly Rate of Decline of Variance HRV LF/HF (All data) | Same as above | SAC |
| 2.120. | FAS | EFF_T1 | Summary of Variance RMSSD (All data) | | SAC |

| Efficacy | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.121. | FAS | EFF_T1 | Summary of Variance RMSSD (Quality data) | | SAC |
| 2.122. | FAS | EFF_T1 | Summary of Change from Baseline of Variance RMSSD (All data) | | SAC |
| 2.123. | FAS | EFF_T1 | Summary of Change from Baseline of Variance RMSSD (Quality data) | | SAC |
| 2.124. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Variance RMSSD (All data) | | SAC |
| 2.125. | FAS | EFF_T1 | Summary of Relative Rate of Variance RMSSD (Quality data) | | SAC |
| 2.126. | FAS | EFF_T1 | Summary of Monthly Rate of Decline of Variance RMSSD (Quality data) | | SAC |
| 2.127. | FAS | EFF_T3 | Statistical Analysis of Relationship between Absolute Values of of HRV endpoints (LF/HF) and Absolute Value of Total ALSFRS-R | | SAC |
| 2.128. | FAS | EFF_T3 | Statistical Analysis of Relationship between Absolute Values of of RMSSD and Absolute Value of Total ALSFRS-R | | SAC |
| 2.129. | FAS | EFF_T3 | Statistical Analysis of Relationship between Change from Baseline of HRV endpoints (LF/HF) and Change from Baseline of Total ALSFRS-R | | SAC |
| 2.130. | FAS | EFF_T3 | Statistical Analysis of Relationship between Change from Baseline of RMSSD and Change from Baseline of Total ALSFRS-R | | SAC |
| 2.131. | FAS | EFF_T3 | Statistical Analysis of Relationship between Slope of HRV endpoints (LF/HF) and Slope of Total ALSFRS-R | | SAC |

| Efficacy | /: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.132. | FAS | EFF_T3 | Statistical Analysis of Relationship between Slope of RMSSD and Slope of Total ALSFRS-R | | SAC |
| Speech | | | | | |
| 2.133. | FAS | EFF_T1 | Summary of Speech Endpoints | Categorise by Test | SAC |
| 2.134. | FAS | EFF_T1 | Summary of Change from Baseline of Speech Endpoints | Categorise by Test | SAC |
| 2.135. | FAS | EFF_T1 | Summary of Relative Rate of Decline of Speech Endpoints | Categorise by Test | SAC |
| 2.136. | FAS | EFF_T1 | Summary of Monthly Rate of Speech Endpoints | Categorise by Test | SAC |
| 2.137. | FAS | EFF_T3 | Statistical Analysis of Relationship between Absolute Values of Speech endpoints and Absolute Value of ALSFRS-R | Paginate by Total Score of ALSFRS,<br>Bulbar Domain and Respiratory Domain | SAC |
| 2.138. | FAS | EFF_T3 | Statistical Analysis of Relationship between Change from Baseline of Speech endpoints and Change from Baseline of ALSFRS-R | Paginate by Total Score of ALSFRS,<br>Bulbar Domain and Respiratory Domain | SAC |
| 2.139. | FAS | EFF_T3 | Statistical Analysis of Relationship between Slope of Speech endpoints and Slope of ALSFRS-R | Paginate by Total Score of ALSFRS,<br>Bulbar Domain and Respiratory Domain | SAC |
| 2.140. | FAS | EFF_T3 | Statistical Analysis of Relationship Absolute Values of Speech endpoints and Absolute Values of FVC | | SAC |
| 2.141. | FAS | EFF_T3 | Statistical Analysis of Relationship between Change from Baseline of Speech endpoints and Change from Baseline of FVC | | SAC |
| 2.142. | FAS | EFF_T3 | Statistical Analysis of Relationship between Slope of Speech endpoints and Slope of FVC | | SAC |
| Data Qu | uality Deviator | | | | |
| 2.143. | FAS | EFF_T2 | Summary of Data Quality Deviators of Actigraphy Data | Footnote the 3 Rules | SAC |
| 2.144. | FAS | EFF_T2 | Summary of Data Quality Deviators of HRV Data | Footnote the 3 Rules | SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Recond | iliation of Action | graphy and Diary | Data | | |
| 2.145. | FAS | EFF_T2 | Summary of Reconciliation of Actigraphy and Diary Data | Footnote: 3 Rules N is the number of subjects at each visit | SAC |
| Actigra | phy Diary – Fe | asibility Measures | 3 | | |
| 2.146. | FAS | EFF_T4 | Summary of Actigraphy Diary (Feasibility) Data | | SAC |
| Device | Impact– Feasil | oility Measures | | | |
| 2.147. | FAS | EFF_T5 | Summary of Device Impact | | SAC |
| ALSFR | S-R | | | | |
| 2.148. | FAS | EFF_T1 | Summary of ALSFRS-R Score | Paginate by Total Score, Gross Motor<br>Domain, Fine Motor Domain, Bulbar<br>Domain and Respiratory Domain | SAC |
| 2.149. | FAS | EFF_T1 | Summary of Change from Baseline of ALSFRS-R Score | Same as Above | SAC |
| 2.150. | FAS | EFF_T1 | Summary of Relative Rate of Decline of ALSFRS-R Score | Same as Above | SAC |
| 2.151. | FAS | EFF_T1 | Summary of Monthly Rate of Decline of ALSFRS-R Score | Same as Above | SAC |
| FVC | | | | | |
| 2.152. | FAS | PD1 | Summary of FVC | | SAC |
| 2.153. | FAS | PD1 | Summary of Change from Baseline of FVC | | SAC |
| 2.154. | FAS | PD1 | Summary of Relative Rate of Decline of FVC | | SAC |
| 2.155. | FAS | PD1 | Summary of Monthly Rate of Decline of FVC | | SAC |

## 9.11.5. Exploratory Figures

| Explora | Exploratory: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Actigra | phy | | | | |
| 2.1. | FAS | EFF_F1 | Plot of Absolute Values of Time Spent Active and Absolute Value of ALSFRS-R v/s Time | Plot Time on X Axis, Endpoint on Y axis and ALSFRS on RHS of Y axis | SAC |
| | | | (All data) | ALSFRS: Total, Fine Motor and Gross<br>Motor | |
| 2.2. | FAS | EFF_F1 | Plot of Absolute Values of Time Spent Active and Absolute Value of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.3. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Time Spent Active and Relative Rate of Decline of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.4. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Time Spent Active and Relative Rate of Decline of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.5. | FAS | EFF_F1 | Plot of Absolute Values of Overall Time Spent Sedentary Not Lying and Absolute Value of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.6. | FAS | EFF_F1 | Plot of Absolute Values of Overall Time Spent Sedentary Not<br>Lying and Absolute Value of ALSFRS-R v/s Time<br>(Quality data) | Same as Above | SAC |
| 2.7. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Overall Time Spent Sedentary<br>Not Lying and Relative Rate of Decline of ALSFRS-R v/s Time<br>(All data) | Same as Above | SAC |

| Explora | Exploratory: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.8. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Overall Time Spent Sedentary<br>Not Lying and Relative Rate of Decline of ALSFRS-R v/s Time<br>(Quality data) | Same as Above | SAC |
| 2.9. | FAS | EFF_F1 | Plot of Absolute Values of Time Spent Lying and Absolute Value of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.10. | FAS | EFF_F1 | Plot of Absolute Values of Time Spent Lying and Absolute Value of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.11. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Time Spent Lying and Relative Rate of Decline of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.12. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Time Spent Lying and Relative Rate of Decline of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.13. | FAS | EFF_F1 | Plot of Absolute Values of Time Spent Sedentary and Absolute Value of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.14. | FAS | EFF_F1 | Plot of Absolute Values of Time Spent Sedentary and Absolute Value of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.15. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Time Spent Sedentary and Relative Rate of Decline of ALSFRS-R v/s Time (All data) | Same as Above | SAC |

| Explora | Exploratory: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.16. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Time Spent Sedentary and Relative Rate of Decline of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.17. | FAS | EFF_F1 | Plot of Absolute Values of Total Activity Score Day/Night and Absolute Value of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.18. | FAS | EFF_F1 | Plot of Absolute Values of Total Activity Score Day/Night and Absolute Value of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.19. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Total Activity Score Day/Night and Relative Rate of Decline of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.20. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Total Activity Score Day/Night and Absolute Value of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.21. | FAS | EFF_F1 | Plot of Absolute Values of Total Activity Score – 24 Hour and Absolute Value of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.22. | FAS | EFF_F1 | Plot of Absolute Values of Total Activity Score – 24 Hour and Absolute Value of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.23. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Total Activity Score – 24 Hour and Relative Rate of Decline of ALSFRS-R v/s Time (All data) | Same as Above | SAC |

| Explora | Exploratory: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.24. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Total Activity Score – 24 Hour and Relative Rate of Decline of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.25. | FAS | EFF_F1 | Plot of Absolute Values of Maximum Score (1 min – 24 Hour Window) and Absolute Value of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.26. | FAS | EFF_F1 | Plot of Absolute Values Maximum Score (1 min – 24 Hour Window) and Absolute Value of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.27. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Maximum Score (1 min – 24 Hour Window) and Relative Rate of Decline of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.28. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Maximum Score (1 min – 24 Hour Window) and Relative Rate of Decline of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.29. | FAS | EFF_F1 | Plot of Absolute Values of Active Periods (Number) and Absolute Value of ALSFRS-R v/s Time (All data) | 5-day time lines (1 for each category) vs ALSFRS on 1 page 5-night time lines vs ALSFRS on 2 <sup>nd</sup> page | SAC |
| 2.30. | FAS | EFF_F1 | Plot of Absolute Values of Active Periods (Number) and Absolute Value of ALSFRS-R v/s Time (Quality data) | 5-day time lines (1 for each category) vs ALSFRS on 1 page 5-night time lines vs ALSFRS on 2 <sup>nd</sup> page | SAC |

| Explora | atory: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.31. | FAS | EFF_F1 | Plot of Active Periods (Number) | Plot of number (y) over time (x) | SAC |
| 2.32. | FAS | EFF_F1 | Plot of Active Periods (Number) and ALSFRS-R v/s Time | 5-day time lines (1 for each category) vs ALSFRS on 1 page 5-night time lines vs ALSFRS on 2 <sup>nd</sup> page | SAC |
| 2.33. | FAS | EFF_F1 | Plot of Absolute Values of Active Periods (Duration) and Absolute Value of ALSFRS-R v/s Time (All data) | Plot Time on X Axis, Endpoint on Y axis and ALSFRS on RHS of Y axis ALSFRS: Total, Fine Motor and Gross Motor | SAC |
| 2.34. | FAS | EFF_F1 | Plot of Absolute Values of Active Periods (Duration) and Absolute Value of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.35. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Active Periods (Duration) and Relative Rate of Decline of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.36. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Active Periods (Duration) and Relative Rate of Decline of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.37. | FAS | EFF_F2 | Scatter Plot of Absolute Values of Actigraphy endpoints and Absolute Value of Total ALSFRS-R | Plot the individual values as dots | SAC |
| 2.38. | FAS | EFF_F2 | Scatter Plot of Change from Baseline of Actigraphy endpoints and Change from Baseline of Total ALSFRS-R | Plot the individual values as dots | SAC |

| Explora | atory: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.39. | FAS | EFF_F2 | Scatter Plot of Slope of Actigraphy endpoints and Slope of Total ALSFRS-R | Plot the individual values as dots | SAC |
| 2.40. | FAS | EFF_F2 | Scatter Plot of Absolute Values of Actigraphy endpoints and Absolute Value of gross motor domain of ALSFRS-R | Plot the individual values as dots | SAC |
| 2.41. | FAS | EFF_F2 | Scatter Plot of Change from Baseline of Actigraphy endpoints and Change from Baseline of gross motor domain of ALSFRS-R | Plot the individual values as dots | SAC |
| 2.42. | FAS | EFF_F2 | Scatter Plot of Slope of Actigraphy endpoints and Slope of gross motor domain of ALSFRS-R | Plot the individual values as dots | SAC |
| 2.43. | FAS | EFF_F2 | Scatter Plot of Absolute Values of Actigraphy endpoints and Absolute Value of fine motor domain of ALSFRS-R | Plot the individual values as dots | SAC |
| 2.44. | FAS | EFF_F2 | Scatter Plot of Change from Baseline of Actigraphy endpoints and Change from Baseline of fine motor domain of ALSFRS-R | Plot the individual values as dots | SAC |
| 2.45. | FAS | EFF_F2 | Scatter Plot of Slope of Actigraphy endpoints and Slope of fine motor domain of ALSFRS-R | Plot the individual values as dots | SAC |
| Night T | ime Rest Endp | oints | | | |
| 2.46. | FAS | EFF_F1 | Plot of Absolute Values of Number Night Time Movement and Absolute Value of ALSFRS-R v/s Time (All data) | Plot Time on X Axis, Endpoint on Y axis and ALSFRS on RHS of Y axis ALSFRS: Total | SAC |
| 2.47. | FAS | EFF_F1 | Plot of Absolute Values of Number Night Time Movement and Absolute Value of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.48. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Number Night Time<br>Movement and Relative Rate of Decline of ALSFRS-R v/s Time<br>(All data) | Same as Above | SAC |

| Explora | Exploratory: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.49. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Number Night Time<br>Movement and Relative Rate of Decline of ALSFRS-R v/s Time<br>(Quality data) | Same as Above | SAC |
| 2.50. | FAS | EFF_F1 | Plot of Absolute Values of Night-time Rest Efficiency and Absolute Value of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.51. | FAS | EFF_F1 | Plot of Absolute Values of Night-time Rest Efficiency and Absolute Value of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.52. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Night-time Rest Efficiency and Relative Rate of Decline of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.53. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Night-time Rest Efficiency and Relative Rate of Decline of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.54. | FAS | EFF_F1 | Plot of Absolute Values of Rest Fragmentation Index and Absolute Value of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.55. | FAS | EFF_F1 | Plot of Absolute Values of Rest Fragmentation Index and Absolute Value of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.56. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Rest Fragmentation Index and Relative Rate of Decline of ALSFRS-R v/s Time (All data) | Same as Above | SAC |

| Exploratory: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.57. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Rest Fragmentation Index and Relative Rate of Decline of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.58. | FAS | EFF_F1 | Plot of Absolute Values of Duration Movement Episodes and Absolute Value of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.59. | FAS | EFF_F1 | Plot of Absolute Values of Duration Movement Episodes and Absolute Value of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.60. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Duration Movement Episodes and Relative Rate of Decline of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.61. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Duration Movement Episodes and Relative Rate of Decline of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.62. | FAS | EFF_F2 | Scatter Plot of Absolute Values of Night Rest Endpoints and Absolute Value of Total ALSFRS-R | Plot the individual values as dots | SAC |
| 2.63. | FAS | EFF_F2 | Scatter Plot of Change from Baseline of Night Rest Endpoints and Change from Baseline of Total ALSFRS-R | Plot the individual values as dots | SAC |
| 2.64. | FAS | EFF_F2 | Scatter Plot of Slope of Night Rest Endpoints and Slope of Total ALSFRS-R | Plot the individual values as dots | SAC |
| Heart F | Rate Variability | | | | |
| 2.65. | FAS | EFF_F1 | Plot of Absolute Values of Mean HRV LF/HF and Absolute Value of ALSFRS-R v/s Time (All data) | Plot Time on X Axis, Endpoint on Y axis and ALSFRS on RHS of Y axis ALSFRS: Total | SAC |

| Explor | Exploratory: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.66. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Mean HRV LF/HF and Relative Rate of Decline of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.67. | FAS | EFF_F1 | Plot of Absolute Values of Mean RMSSD and Absolute Value of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.68. | FAS | EFF_F1 | Plot of Absolute Values of Mean RMSSD and Absolute Value of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.69. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Mean RMSSD and Relative Rate of Decline of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.70. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Mean RMSSD and Relative Rate of Decline of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.71. | FAS | EFF_F1 | Plot of Absolute Values of Variance HRV LF/HF and Absolute Value of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.72. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Variance HRV LF/HF and Relative Rate of Decline of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.73. | FAS | EFF_F1 | Plot of Absolute Values of Variance RMSSD and Absolute Value of ALSFRS-R v/s Time (All data) | Same as Above | SAC |

| Exploratory: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.74. | FAS | EFF_F1 | Plot of Absolute Values of Variance RMSSD and Absolute Value of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.75. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Variance RMSSD and Relative Rate of Decline of ALSFRS-R v/s Time (All data) | Same as Above | SAC |
| 2.76. | FAS | EFF_F1 | Plot of Relative Rate of Decline of Variance RMSSD and Relative Rate of Decline of ALSFRS-R v/s Time (Quality data) | Same as Above | SAC |
| 2.77. | FAS | EFF_F2 | Scatter Plot of Absolute Values of HRV endpoints (LF/HF) and Absolute Value of Total ALSFRS-R | Plot individual values as dots | SAC |
| 2.78. | FAS | EFF_F2 | Scatter Plot of Absolute Values of RMSSD and Absolute Value of Total ALSFRS-R | Plot individual values as dots | SAC |
| 2.79. | FAS | EFF_F2 | Scatter Plot of Change from Baseline of HRV endpoints (LF/HF) and Change from Baseline of Total ALSFRS-R | Plot individual values as dots | SAC |
| 2.80. | FAS | EFF_F2 | Scatter Plot of Change from Baseline of RMSSD and Change from Baseline of Total ALSFRS-R | Plot individual values as dots | SAC |
| 2.81. | FAS | EFF_F2 | Scatter Plot of Slope of HRV endpoints (LF/HF) and Slope of Total ALSFRS-R | Plot individual values as dots | SAC |
| 2.82. | FAS | EFF_F2 | Scatter Plot of Slope of RMSSD and Slope of Total ALSFRS-R | Plot individual values as dots | SAC |
| Speech | i | | | | |
| 2.83. | FAS | EFF_F1 | Plot of Absolute Values of Speech Endpoints and Absolute Values of ALSFRS-R v/s Time | Plot Time on X Axis, Endpoint on Y axis and ALSFRS on RHS of Y axis ALSFRS: Total Bulbar and Respiratory Domain | SAC |

| Explora | atory: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.84. | FAS | EFF_F1 | Plot of Relative Rate of decline of Speech Endpoints and Relative Rate of decline of ALSFRS-R v/s Time | Same as Above | SAC |
| 2.85. | FAS | EFF_F2 | Scatter Plot of Absolute Values of Speech endpoints and Absolute Value of ALSFRS-R | Plot individual values as dots | SAC |
| 2.86. | FAS | EFF_F2 | Scatter Plot of Change from Baseline of Speech endpoints and Change from Baseline of ALSFRS-R | Plot individual values as dots | SAC |
| 2.87. | FAS | EFF_F2 | Scatter Plot of Slope of Speech endpoints and Slope of ALSFRS-R | Plot individual values as dots | SAC |
| 2.88. | FAS | EFF_F2 | Scatter Plot of Absolute Values of Speech endpoints and Absolute Values of FVC | Plot individual values as dots | SAC |
| 2.89. | FAS | EFF_F2 | Scatter Plot of Change from Baseline of Speech endpoints and Change from Baseline of FVC | Plot individual values as dots | SAC |
| 2.90. | FAS | EFF_F2 | Scatter Plot of Slope of Speech endpoints and Slope of FVC | Plot individual values as dots | SAC |
| ALSFR | S-R | | | | |
| 2.91. | FAS | EFF_F1 | Mean (SE) Plot of ALSFRS-R Score | <ul> <li>Paginate by Total Score,<br/>Gross Motor Domain, Fine<br/>Motor Domain, Bulbar<br/>Domain and Respiratory<br/>Domain</li> <li>Only 1 y axis</li> </ul> | SAC |
| 2.92. | FAS | EFF_F1 | Mean (SE) Plot of Relative Rate of Decline of ALSFRS-R Score | <ul> <li>Paginate by Total Score,<br/>Gross Motor Domain, Fine<br/>Motor Domain, Bulbar<br/>Domain and Respiratory<br/>Domain</li> <li>Only 1 y axis</li> </ul> | SAC |

| Exploratory: Figures | | | | | |
|---|---|---|---|---|---|
| No. | No. Population IDSL / TST ID / Example Shell Title Programming Notes Delive [Prior | | | | |
| FVC | | | | | |
| 2.93. | FAS | EFF_F1 | Mean (SE) Plot of FVC | Only 1 y axis | SAC |
| 2.94. | FAS | EFF_F1 | Mean (SE) Plot of Relative Rate of FVC | Same as above | SAC |

### 9.11.6. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 3.1. | Safety | AE1CP | Summary of All Adverse Events | Add a Footnote: Only those AEs and SAEs which, in the opinion of the investigator, are related to a protocol-mandated procedure or one of the devices used in the study will be reported | SAC |
| 3.2. | Safety | AE1CP | Summary of Serious Adverse Events | | SAC |
| 3.3. | Safety | AE1CP | Summary of Adverse Events Leading to Withdrawal from Study | | SAC |
| 3.4. | Safety | AE5A | Summary of Adverse Events by Maximum Intensity | | SAC |
| 3.5. | Safety | SAFE_T1 | Summary of Deaths | | SAC |

## 9.11.7. ICH Listings

| ICH : L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | Screen<br>Failure | ES7 | Listing of Reasons for Screen Failure | | SAC |
| 2. | FAS | ES2 | Listing of Reasons for Study Withdrawal | | SAC |
| Protoc | ol Deviations | | | | · |
| 3. | FAS | DV2 | Listing of Important Protocol Deviations | | SAC |
| 4. | FAS | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC |
| Popula | tions Analysed | | | | |
| 5. | Enrolled | SA3a | Listing of Subjects Excluded from Any Population | | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 6. | FAS | DM2 | Listing of Demographic Characteristics | | SAC |
| 7. | FAS | DM10 | Listing of Race | | SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 8. | FAS | MH3 | Listing of Medical Conditions | | SAC |
| 9. | FAS | CP_CM3 | Listing of Concomitant Medications | | SAC |
| Advers | se Events | | | | |
| 10. | Safety | CP_AE8 | Listing of All Adverse Events | | SAC |
| 11. | Safety | CP_AE8 | Listing of Drug Related Adverse Events | | SAC |
| 12. | Safety | CP_AE8 | Listing of Serious Adverse Events | | SAC |
| 13. | Safety | CP_AE8 | Listing of Adverse Events Leading to Withdrawal from Study | | SAC |

| ICH : Li | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 14. | Safety | CP_AE8 | Listing of Adverse Events by Maximum Intensity | | SAC |
| Death | Death | | | | |
| 15. | Safety | SAFE_L1 | Listing of Deaths | | SAC |

## 9.11.8. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | se Events | | | | |
| 16. | Safety | AE2 | Listing of Relationship between System Organ Class and Verbatim Text | | SAC |
| Actigra | phy | | | | |
| 17. | FAS | PD11 | Listing of Wear Time - Derived Data (All data) | | SAC |
| 18. | FAS | PD11 | Listing of Wear Time - Derived Data (Quality Data data) | | SAC |
| 19. | FAS | PD11 | Listing of Duration of Day Time Wear Time (All data) | | SAC |
| 20. | FAS | PD11 | Listing of Duration of Day Time Wear Time (Quality data) | | SAC |
| 21. | FAS | PD11 | Listing of Duration of Night Time Wear Time (All data) | | SAC |
| 22. | FAS | PD11 | Listing of Duration of Night Time Wear Time (Quality data) | | SAC |
| 23. | FAS | PD11 | Listing of Time Spent Active – Raw Data | | SAC |
| 24. | FAS | PD11 | Listing of Time Spent Active – Derived Data (All data) | | SAC |
| 25. | FAS | PD11 | Listing of Time Spent Active – Derived Data (Quality data) | | SAC |
| 26. | FAS | PD11 | Listing of Over All Time Spent sedentary not Lying – Raw Data | | SAC |

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 27. | FAS | PD11 | Listing of Over All Time Spent sedentary not Lying – Derived Data (All data) | | SAC |
| 28. | FAS | PD11 | Listing of Over All Time Spent sedentary not Lying – Derived Data (Quality data) | | SAC |
| 29. | FAS | PD11 | Listing of Over All Time Spent Lying – Raw Data | | SAC |
| 30. | FAS | PD11 | Listing of Over All Time Spent Lying – Derived Data (All data) | | SAC |
| 31. | FAS | PD11 | Listing of Over All Time Spent Lying – Derived Data (Quality data) | | SAC |
| 32. | FAS | PD11 | Listing of Over All Time Spent Sedentary – Raw Data | | SAC |
| 33. | FAS | PD11 | Listing of Over All Time Spent Sedentary – Derived Data (All data) | | SAC |
| 34. | FAS | PD11 | Listing of Over All Time Spent Sedentary – Derived Data (Quality data) | | SAC |
| 35. | FAS | PD11 | Listing of Total Activity Score Day/Night – Raw Data | | SAC |
| 36. | FAS | PD11 | Listing of Total Activity Score Day/Night – Derived Data (All data) | | SAC |
| 37. | FAS | PD11 | Listing of Total Activity Score Day/Night – Derived Data (Quality data) | | SAC |
| 38. | FAS | PD11 | Listing of Total Activity Score – 24 Hour – Raw Data | | SAC |

| Non-ICH : Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 39. | FAS | PD11 | Listing of Total Activity Score – 24 Hour – Derived Data (All data) | | SAC |
| 40. | FAS | PD11 | Listing of Total Activity Score – 24 Hour – Derived Data (Quality data) | | SAC |
| 41. | FAS | PD11 | Listing of Maximum Score from 1 – 24 Hour Window -Raw Data | | SAC |
| 42. | FAS | PD11 | Listing of Maximum Score from 1 – 24 Hour Window - Derived Data (All data) | | SAC |
| 43. | FAS | PD11 | Listing of Maximum Score from 1 – 24 Hour Window - Derived Data (Quality data) | | SAC |
| 44. | FAS | PD11 | Listing of Active Periods (Numbers) – Raw Data | | SAC |
| 45. | FAS | PD11 | Listing of Active Periods (Numbers) – Derived Data (All data) | | SAC |
| 46. | FAS | PD11 | Listing of Active Periods (Numbers) – Derived Data (Quality data) | | SAC |
| 47. | FAS | PD11 | Listing of Active Periods (Duration) – Raw Data | | SAC |
| 48. | FAS | PD11 | Listing of Active Periods (Duration) – Derived Data (All data) | | SAC |
| 49. | FAS | PD11 | Listing of Active Periods (Duration) – Derived Data (Quality data) | | SAC |

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Night T | ime Rest Endp | oints | | | <u> </u> |
| 50. | FAS | PD11 | Listing of Number Night Time Movement Episodes/Hr (All data) | | SAC |
| 51. | FAS | PD11 | Listing of Number Night Time Movement Episodes/Hr (Quality data) | | SAC |
| 52. | FAS | PD11 | Listing of Percent Time Night-time Rest Efficiency (All data) | | SAC |
| 53. | FAS | PD11 | Listing of Percent Time Night-time Rest Efficiency (Quality data) | | SAC |
| 54. | FAS | PD11 | Listing of Rest Fragmentation Index (All data) | | SAC |
| 55. | FAS | PD11 | Listing of Rest Fragmentation Index (Quality data) | | SAC |
| 56. | FAS | PD11 | Listing of Average Duration Movement Episodes (All data) | | SAC |
| 57. | FAS | PD11 | Listing of Average Duration Movement Episodes (Quality data) | | SAC |
| Heart F | Rate Variability | 1 | | | 1 |
| 58. | FAS | PD11 | Listing of Mean HRV LF/HF (All data) | | SAC |
| 59. | FAS | PD11 | Listing of Mean RMSSD (All data) | | SAC |
| 60. | FAS | PD11 | Listing of Mean RMSSD (Quality data) | | SAC |
| 61. | FAS | PD11 | Listing of Variance HRV LF/HF (All data) | | SAC |
| 62. | FAS | PD11 | Listing of Variance RMSSD (All data) | | SAC |

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 63. | FAS | PD11 | Listing of Variance RMSSD (Quality data) | | SAC |
| 64. | FAS | PD11 | Listing of HRV data from McLaren | | SAC |
| Speech | 1 | | | | |
| 65. | FAS | PD11 | Listing of Speech Endpoints | Also include comments | SAC |
| Actigra | phy Diary Data | | | | |
| 66. | FAS | PD11 | Listing of Actigraphy Diary (Feasibility) Data | For categorical data add the test and the categorical results | SAC |
| Device | Impact | | | | |
| 67. | FAS | PD11 | Listing of Device Impact | For categorical data add the test and the categorical results | SAC |
| Neurol | ogical Exam | | | | |
| 68. | FAS | PD11 | Listing of Neurological Exams | For categorical data add the test and the categorical results, add location and laterality | |
| ALSFR | S-R | | | | |
| 69. | FAS | PD11 | Listing of ALSFRS-R | | SAC |
| FVC | • | | | | |
| 70. | FAS | PD11 | Listing of FVC | | SAC |